CLINICAL TRIAL: NCT02344290
Title: Randomized Trial to Prevent Vascular Events in HIV - REPRIEVE
Brief Title: Evaluating the Use of Pitavastatin to Reduce the Risk of Cardiovascular Disease in HIV-Infected Adults
Acronym: REPRIEVE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); Kowa Pharmaceuticals America, Inc. (Industry); Gilead Sciences (Industry); Massachusetts General Hospital (Other); NEAT ID Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: A5332; 11960 (Other: DAIDS-ES Registry Number); 1U01HL123339-01 (NIH); 1U01HL123336-01 (NIH); EU5332 (Other: Massachusetts General Hospital)
Record Dates: First submitted 2015-01-16; First posted 2015-01-22 (Estimated); Results first posted 2024-10-15 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-09

CONDITIONS: HIV; Cardiovascular Diseases
Keywords: HIV; Cardiovascular Disease; Myocardial Infarction; Inflammation; Statin; Computerized Tomography; Cholesterol; COVID-19
MeSH Terms: conditions — Cardiovascular Diseases; Myocardial Infarction; Inflammation; COVID-19 | interventions — pitavastatin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Pitavastatin (Experimental): Participants received pitavastatin once a day for the entire time they were in study follow-up.
  Interventions: Drug: Pitavastatin
- Placebo (Placebo Comparator): Participants received placebo for pitavastatin once a day for the entire time they were in study follow-up.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Pitavastatin — One tablet (4 mg) taken once daily, orally with or without food
  Arms: Pitavastatin
Drug: Placebo — One tablet taken once daily, orally with or without food
  Arms: Placebo

SUMMARY:
People with HIV are at risk for cardiovascular disease (CVD). This study evaluated the use of pitavastatin to reduce the risk of CVD in adults with HIV on antiretroviral therapy (ART).

The REPRIEVE trial consisted of two parallel identical protocols:

* REPRIEVE (A5332) was funded by the NHLBI, with additional infrastructure support provided by the NIAID, and was conducted in U.S and select international sites (approximately 120 sites in 11 countries).
* REPRIEVE (EU5332) was co-sponsored by NEAT ID and MGH, and was conducted at 13 sites in Spain.

DETAILED DESCRIPTION:
There are few strategies to prevent CVD in people with HIV (PWH), even though they are at high risk for developing CVD. Statin medications are used to lower cholesterol and may be effective at reducing the risk of CVD in PWH. The purpose of this study was to evaluate the use of pitavastatin to reduce the risk of CVD in PWH on ART.

This study enrolled PWH who were on any ART regimen (ART was not provided by the study) for at least 6 months before study entry and were at low to moderate risk of CVD using the 2013 American College of Cardiology (ACC)/American Heart Association (AHA) guideline thresholds for recommended statin initiation.

Participants were randomly assigned to receive 4 mg of pitavastatin or placebo once a day for their entire study duration. Pitavastatin or placebo could be discontinued and clinically indicated statin therapy initiated at the discretion of the site investigator or the participant's care provider, with the intention of following the participant according to the intention-to-treat trial design. Study visits occurred at study entry and Months 1 and 4. Starting at Month 4, study visits occurred every 4 months for the rest of the study. Depending on when participants enrolled, they were in the study for a total of 4 to 8 years. Study visits included medical and medication history reviews, physical examinations, blood collections, assessments and questionnaires, urine collections (for some participants), and an electrocardiogram (ECG) (at study entry only).

Participants at US sites had the option of enrolling in a substudy (Effects of Pitavastatin on Coronary Artery Disease and Inflammatory Biomarkers: Mechanistic Substudy of REPRIEVE [A5333s]). The substudy evaluated the effect of pitavastatin on the progression of non-calcified coronary atherosclerotic plaque (NCP) and inflammatory biomarkers in PWH. Participants in the substudy attended study visits at study entry and Months 4 and 24. The visits included questionnaires and assessments, a blood collection, and a coronary computed tomography angiography (CCTA). The Mechanistic Substudy closed to accrual on February 6, 2018, when its accrual target of 800 participants had been reached. Sites that enrolled participants into the Mechanistic Substudy are indicated with asterisk (*) at the end of the institution names in the Contacts and Locations section.

Participants enrolled in REPRIEVE from select study sites, including international sites, through December, 2017, were included in the REPRIEVE Kidney Function Objectives Cohort to evaluate the effects of pitavastatin on parameters of kidney function in the setting of HIV. These objectives include evaluating high risk groups and mechanisms driving kidney function decline in the setting of HIV.

Women and men enrolled in REPRIEVE after February, 2016 were included in an observational cohort (REPRIEVE Women's Objectives Cohort) facilitating assessment of sex-specific mechanisms of CVD risk and risk reduction among PWH. This effort also included an evidence-based recruitment campaign to enhance women's participation in REPRIEVE.

In response to the SARS-CoV-2 pandemic, a supplemental objective was added in 2020. To better understand how COVID-19 affects PWH and if pitavastatin may reduce the risk of serious COVID-19 disease, we evaluated interrelated but independent key topics including epidemiology, host factors, and protective strategies. Starting from April 2020, COVID-19 assessment was completed at each study visit, and blood was collected for COVID-19 biomarkers.

The data and safety monitoring board (DSMB) recommended stopping the trial for efficacy at the second planned review on March 30, 2023, and concluded that no unexpected safety concerns had been reported. Following the DSMB action, participants were asked to return for the final study visit. All final visits were completed by August 21, 2023. We here present the results based on the final trial database, including the full follow-up out to closeout visits.

ELIGIBILITY:
Inclusion Criteria:

* Individual with HIV-1
* Combination antiretroviral therapy (ART) for at least 180 days prior to study entry
* CD4+ cell count greater than 100 cells/mm^3
* Acceptable screening laboratories including:

  * Fasting low-density lipoprotein (LDL) cholesterol as follows:

    * If ASCVD risk score was less than 7.5%, LDL cholesterol must have been less than 190 mg/dL.
    * If ASCVD risk score was greater than or equal to 7.5% and less than or equal to 10%, LDL must have been less than 160 mg/dL.
    * If ASCVD risk score was greater than 10% and less than or equal to 15%, LDL must have been less than 130 mg/dL.
    * Participants with LDL less than 70 mg/dL were eligible regardless of the 10-year ASCVD risk score, in line with the ACC/AHA 2013 Prevention Guidelines.
  * Fasting triglycerides less than 500 mg/dL
  * Hemoglobin greater than or equal to 8 g/dL for female participants and greater than or equal to 9 g/dL for male participants
  * Glomerular filtration rate (GFR) greater than or equal to 60 mL/min/1.73m^2 or creatinine clearance (CrCl) greater than or equal to 60 mL/min
  * Alanine aminotransferase (ALT) less than or equal to 2.5 x the upper limit of normal (ULN)
* For persons with known chronic active hepatitis B or C, calculated fibrosis 4 score (FIB-4) must have been less than or equal to 3.25
* Ability and willingness of participant or legal representative to provide written informed consent

Exclusion Criteria:

* Clinical ASCVD, as defined by 2013 American College of Cardiology (ACC)/American Heart Association (AHA) guidelines, including a previous diagnosis of any of the following:

  * Acute myocardial infarction (AMI)
  * Acute coronary syndromes
  * Stable or unstable angina
  * Coronary or other arterial revascularization
  * Stroke
  * Transient ischemic attack (TIA)
  * Peripheral arterial disease presumed to be of atherosclerotic origin
* Current diabetes mellitus with LDL greater than or equal to 70 mg/dL
* 10-year ASCVD risk score estimated by Pooled Cohort Equations greater than 15%
* Active cancer within 12 months prior to study entry, except successfully treated non-melanomatous skin cancer and Kaposi sarcoma without visceral organ involvement
* Known decompensated cirrhosis
* History of myositis or myopathy with active disease in the 180 days prior to study entry
* Known untreated symptomatic thyroid disease
* History of allergy or severe adverse reaction to statins
* Use of specific immunosuppressants or immunomodulatory agents including but not limited to tacrolimus, sirolimus, rapamycin, mycophenolate, cyclosporine, tumor necrosis factor (TNF)-alpha blockers or antagonists, azathioprine, interferon, growth factors, or intravenous immunoglobulin (IVIG) in the 30 days prior to study entry.
* Current use of erythromycin, colchicine, or rifampin
* Use of any statin drugs, gemfibrozil, or PCSK9 inhibitors in the 90 days prior to study entry
* Current use of an investigational new drug that would be contraindicated
* Serious illness or trauma requiring systemic treatment or hospitalization in the 30 days prior to study entry
* Current pregnancy or breastfeeding
* Alcohol or drug use that, in the opinion of the site investigator, would interfere with completion of study procedures
* Other medical, psychiatric, or psychological condition that, in the opinion of the site investigator, would interfere with completion of study procedures and or adherence to study drug

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7769 (Actual)
Dates: Start 2015-03-26 (Actual); Primary Completion 2023-08-21 (Actual); Study Completion 2023-08-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven Grinspoon, MD, Study Chair — Harvard Medical School (HMS and HSDM)
Locations (137):
- United States (91):
  - Alabama CRS*, Birmingham, Alabama
  - University of Arizona CRS, Tucson, Arizona
  - University of Southern California CRS*, Los Angeles, California
  - UCLA CARE Center CRS*, Los Angeles, California
  - Mills Clinical Research CRS, Los Angeles, California
  - VA West Los Angeles Medical Center CRS, Los Angeles, California
  - Los Angeles LGBT Center CRS, Los Angeles, California
  - Eisenhower Health Center at Rimrock CRS, Palm Springs, California
  - Stanford AIDS Clinical Trials Unit CRS, Palo Alto, California
  - UCSD Antiviral Research Center CRS*, San Diego, California
  - Ucsf Hiv/Aids Crs*, San Francisco, California
  - Harbor-UCLA CRS*, Torrance, California
  - University of Colorado Hospital CRS*, Aurora, Colorado
  - Denver Public Health CRS, Denver, Colorado
  - Yale University CRS, New Haven, Connecticut
  - VA Connecticut Healthcare System CRS, West Haven, Connecticut
  - Whitman-Walker Health CRS, Washington D.C., District of Columbia
  - Georgetown University CRS (GU CRS), Washington D.C., District of Columbia
  - Capital Medical Associates, PC CRS, Washington D.C., District of Columbia
  - Infectious Diseases Clinic, Washington DC Veterans Affairs Medical Center CRS, Washington D.C., District of Columbia
  - Malcom Randall VA Medical Center CRS, Gainesville, Florida
  - AHF-The Kinder Medical Group CRS, Miami, Florida
  - The University of Miami AIDS Clinical Research Unit (ACRU) CRS, Miami, Florida
  - University of Miami Infectious Disease Research Unit at Jackson Memorial Hospital CRS, Miami, Florida
  - AHF - South Beach CRS, Miami, Florida
  - Orlando Immunology Center CRS, Orlando, Florida
  - Community AIDS Network/Comprehensive Care Clinic CRS, Sarasota, Florida
  - Florida Department of Health - Hillsborough County, Tampa, Florida
  - AIDS Research and Treatment Center of the Treasure Coast CRS, Vero Beach, Florida
  - The Ponce de Leon Center CRS, Atlanta, Georgia
  - Augusta University Research Institute, Inc. CRS, Augusta, Georgia
  - Northwestern University CRS*, Chicago, Illinois
  - Rush University CRS*, Chicago, Illinois
  - UIC Project WISH CRS, Chicago, Illinois
  - Indiana University Infectious Diseases Research CRS, Indianapolis, Indiana
  - Department of Internal Medicine, University of Iowa Hospitals & Clinics CRS, Iowa City, Iowa
  - Bluegrass Care Clinic/University of Kentucky Research Foundation CRS, Lexington, Kentucky
  - 550 Clinic -University of Louisville CRS, Louisville, Kentucky
  - Tulane - Louisiana Community AIDS Research Program (T-LaCARP) CRS, New Orleans, Louisiana
  - Johns Hopkins University CRS*, Baltimore, Maryland
  - Tufts Medical Center CRS, Boston, Massachusetts
  - Massachusetts General Hospital CRS (MGH CRS)*, Boston, Massachusetts
  - Brigham and Women's Hospital Therapeutics Clinical Research Site (BWH TCRS) CRS*, Boston, Massachusetts
  - Boston Medical Center CRS, Boston, Massachusetts
  - Baystate Infectious Diseases Clinical Research CRS, Springfield, Massachusetts
  - Henry Ford Hosp. CRS, Detroit, Michigan
  - St. John Newland Medical Associates CRS, Southfield, Michigan
  - Abbott Northwestern Hospital CRS, Minneapolis, Minnesota
  - University of Mississippi Medical Center CRS, Jackson, Mississippi
  - Washington University Therapeutics (WT) CRS*, St Louis, Missouri
  - Specialty Care Center CRS, Omaha, Nebraska
  - Cooper Univ. Hosp. CRS, Camden, New Jersey
  - New Jersey Medical School Clinical Research Center CRS*, Newark, New Jersey
  - Mount Sinai Beth Israel CRS*, New York, New York
  - VA New York Harbor Healthcare System (NYHHS), NY Campus CRS, New York, New York
  - Weill Cornell Chelsea CRS*, New York, New York
  - Mount Sinai Downtown CRS*, New York, New York
  - Mount Sinai West Samuels CRS*, New York, New York
  - Mount Sinai St. Luke's Morningside CRS*, New York, New York
  - Infectious Disease Clinical and Translational Research Center (CTRC) CRS, New York, New York
  - Columbia P&S CRS*, New York, New York
  - Weill Cornell Uptown CRS*, New York, New York
  - University of Rochester Adult HIV Therapeutic Strategies Network CRS*, Rochester, New York
  - James J Peters VA Medical Center CRS, The Bronx, New York
  - Chapel Hill CRS*, Chapel Hill, North Carolina
  - Duke University Medical Center CRS, Durham, North Carolina
  - Greensboro CRS*, Greensboro, North Carolina
  - Wake Forest Baptist Medical Center CRS, Winston-Salem, North Carolina
  - Cincinnati Clinical Research Site*, Cincinnati, Ohio
  - Case Clinical Research Site*, Cleveland, Ohio
  - Ohio State University CRS*, Columbus, Ohio
  - University of Toledo Medical Center CRS, Toledo, Ohio
  - Oklahoma State University Center for Health Sciences CRS, Tulsa, Oklahoma
  - Division of Infectious Diseases Clinical Research Center- Drexel University CRS, Philadelphia, Pennsylvania
  - Penn Therapeutics, CRS*, Philadelphia, Pennsylvania
  - Center of Translational AIDS Research, Lewis Katz School of Medicine at Temple University CRS, Philadelphia, Pennsylvania
  - Positive Health Clinic CRS, Pittsburgh, Pennsylvania
  - University of Pittsburgh CRS*, Pittsburgh, Pennsylvania
  - The Miriam Hospital Clinical Research Site (TMH CRS) CRS*, Providence, Rhode Island
  - Medical University of South Carolina: Division of Infectious Diseases CRS, Charleston, South Carolina
  - Prisma Health CRS, Columbia, South Carolina
  - Vanderbilt Therapeutics (VT) CRS*, Nashville, Tennessee
  - Trinity Health and Wellness Center CRS, Dallas, Texas
  - Dallas VA Medical Center CRS, Dallas, Texas
  - UT Southwestern HIV/ID Clinical Trials Unit CRS, Dallas, Texas
  - Houston AIDS Research Team CRS*, Houston, Texas
  - Michael E. DeBakey VAMC REPRIEVE CRS, Houston, Texas
  - Inova Heart and Vascular Institute CRS, Falls Church, Virginia
  - Virginia Commonwealth University CRS, Richmond, Virginia
  - University of Washington AIDS CRS*, Seattle, Washington
  - Medical College of Wisconsin, Inc. CRS, Milwaukee, Wisconsin
- Gaborone CRS, Gaborone, South-East District, Botswana
- Brazil (10):
  - Tropical Medicine Foundation Dr. Heitor Vieira Dourado CRS, Manaus, Amazonas
  - School of Medicine, Federal University of Minas Gerais CRS, Belo Horizonte, Minas Gerais
  - HGNI HIV Family Care Clinic - HHFCC CRS, Nova Iguaçu, Rio de Janeiro
  - Hospital Nossa Senhora da Conceicao CRS, Porto Alegre, Rio Grande do Sul
  - Centro de Referencia e Treinamento DST/AIDS CRS, São Paulo, São Paulo
  - Projeto Praça Onze Pesquisa em Saúde CRS, Rio de Janeiro
  - Hospital Federal dos Servidores do Estado CRS, Rio de Janeiro
  - Instituto de Pesquisa Clinica Evandro Chagas (IPEC) CRS, Rio de Janeiro
  - Instituto de Infectologia Emilio Ribas CRS, São Paulo
  - Centro de Pesquisas Clínicas IC-HCFMUSP CRS, São Paulo
- Canada (6):
  - Vancouver ID Research & Care Centre Society CRS, Vancouver, British Columbia
  - Hamilton Health Sciences - Special Immunology Services Clinic CRS, Hamilton, Ontario
  - Maple Leaf Research CRS, Toronto, Ontario
  - Toronto General Hospital CRS, Toronto, Ontario
  - Chronic Viral Illness Service CRS, Montreal, Quebec
  - Centre hospitalier de l'Université Laval CRS, Québec, Quebec
- Haiti (2):
  - GHESKIO Institute of Infectious Diseases and Reproductive Health (GHESKIO - IMIS) CRS, Port-au-Prince
  - Les Centres GHESKIO Clinical Research Site (GHESKIO-INLR) CRS, Port-au-Prince
- India (2):
  - Byramjee Jeejeebhoy Medical College (BJMC) CRS, Pune, Maharashtra
  - Chennai Antiviral Research and Treatment (CART) CRS, Chennai, Tamil Nadu
- Peru (2):
  - Barranco CRS, Lima
  - San Miguel CRS, Lima
- Puerto Rico AIDS Clinical Trials Unit CRS*, San Juan, PR, Puerto Rico
- South Africa (5):
  - Soweto ACTG CRS, Johannesburg, Gauteng
  - Wits Helen Joseph Hospital CRS (Wits HJH CRS), Johannesburg, Gauteng
  - Durban International Clinical Research Site CRS, Durban, KwaZulu-Natal
  - University of Cape Town Lung Institute (UCTLI) CRS, Cape Town, Western Cape
  - Famcru Crs, Tygerberg, Western Cape
- Spain (13):
  - Hospital General Universitario de Alicante, Alicante
  - Hospital Germans Trias i Pujol, Badalona
  - Hospital Universitario Valle d'Hebron, Barcelona
  - Hospital Clinic de Barcelona, Barcelona
  - Hospital Universitario de Bellvitge, Barcelona
  - Hospital Universitario de Basurto de Basurto, Bilbao
  - Hospital General Universitario De Elche, Elche
  - Hospital Gregorio Universitario Maranon, Madrid
  - Hospital Universitario Ramon y Cajal, Madrid
  - Hospital Universitario Clinico San Carlos, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitario Virgen de la Victoria, Málaga
- Thailand (2):
  - Thai Red Cross AIDS Research Centre (TRC-ARC) CRS, Bangkok
  - Chiang Mai University HIV Treatment (CMU HIV Treatment) CRS, Chiang Mai
- Joint Clinical Research Centre (JCRC)/Kampala Clinical Research Site, Kampala, Uganda
- Milton Park CRS, Harare, Zimbabwe

REFERENCES:
- [Background] Goff DC Jr, Lloyd-Jones DM, Bennett G, Coady S, D'Agostino RB Sr, Gibbons R, Greenland P, Lackland DT, Levy D, O'Donnell CJ, Robinson JG, Schwartz JS, Shero ST, Smith SC Jr, Sorlie P, Stone NJ, Wilson PWF. 2013 ACC/AHA guideline on the assessment of cardiovascular risk: a report of the American College of Cardiology/American Heart Association Task Force on Practice Guidelines. J Am Coll Cardiol. 2014 Jul 1;63(25 Pt B):2935-2959. doi: 10.1016/j.jacc.2013.11.005. Epub 2013 Nov 12. No abstract available. PMID 24239921
- [Result] Zanni MV, Fitch K, Rivard C, Sanchez L, Douglas PS, Grinspoon S, Smeaton L, Currier JS, Looby SE. Follow YOUR Heart: development of an evidence-based campaign empowering older women with HIV to participate in a large-scale cardiovascular disease prevention trial. HIV Clin Trials. 2017 Mar;18(2):83-91. doi: 10.1080/15284336.2017.1297551. PMID 28277924
- [Result] Grinspoon SK, Fitch KV, Overton ET, Fichtenbaum CJ, Zanni MV, Aberg JA, Malvestutto C, Lu MT, Currier JS, Sponseller CA, Waclawiw M, Alston-Smith B, Cooper-Arnold K, Klingman KL, Desvigne-Nickens P, Hoffmann U, Ribaudo HJ, Douglas PS; REPRIEVE Investigators. Rationale and design of the Randomized Trial to Prevent Vascular Events in HIV (REPRIEVE). Am Heart J. 2019 Jun;212:23-35. doi: 10.1016/j.ahj.2018.12.016. Epub 2019 Mar 4. PMID 30928825
- [Result] Hoffmann U, Lu MT, Olalere D, Adami EC, Osborne MT, Ivanov A, Aluru JS, Lee S, Arifovic N, Overton ET, Fichtenbaum CJ, Aberg JA, Alston-Smith B, Klingman KL, Waclawiw M, Burdo TH, Williams KC, Zanni MV, Desvigne-Nickens P, Cooper-Arnold K, Fitch KV, Ribaudo H, Douglas PS, Grinspoon SK; REPRIEVE Investigators. Rationale and design of the Mechanistic Substudy of the Randomized Trial to Prevent Vascular Events in HIV (REPRIEVE): Effects of pitavastatin on coronary artery disease and inflammatory biomarkers. Am Heart J. 2019 Jun;212:1-12. doi: 10.1016/j.ahj.2019.02.011. Epub 2019 Mar 4. PMID 30928823
- [Result] Grinspoon SK, Douglas PS, Hoffmann U, Ribaudo HJ. Leveraging a Landmark Trial of Primary Cardiovascular Disease Prevention in Human Immunodeficiency Virus: Introduction From the REPRIEVE Coprincipal Investigators. J Infect Dis. 2020 Jul 9;222(Suppl 1):S1-S7. doi: 10.1093/infdis/jiaa098. PMID 32645161
- [Result] Fitch KV, Kileel EM, Looby SE, Zanni MV, Sanchez LR, Fichtenbaum CJ, Overton ET, Malvestutto C, Aberg JA, Klingman KL, Alston-Smith B, Lavelle J, Rancourt A, Badal-Faesen S, Cardoso SW, Avihingsanon A, Patil S, Sponseller CA, Melbourne K, Ribaudo HJ, Cooper-Arnold K, Desvigne-Nickens P, Hoffmann U, Douglas PS, Grinspoon SK; REPRIEVE Investigators. Successful recruitment of a multi-site international randomized placebo-controlled trial in people with HIV with attention to diversity of race and ethnicity: critical role of central coordination. HIV Res Clin Pract. 2020 Feb;21(1):11-23. doi: 10.1080/25787489.2020.1733794. Epub 2020 Mar 11. PMID 32160827
- [Result] Overton ET, Kantor A, Fitch KV, Muntner P, Supparatpinyo K, Mosepele M, Mohapi L, Cardoso SW, Patil S, de Lacerda MVG, McComsey G, Aberg JA, Douglas PS, Grinspoon SK, Ribaudo H, Wyatt CM. An Evaluation of Baseline Kidney Function in the REPRIEVE Trial of Pitavastatin in Human Immunodeficiency Virus. J Infect Dis. 2020 Jul 9;222(Suppl 1):S41-S51. doi: 10.1093/infdis/jiaa222. PMID 32645164
- [Result] Fichtenbaum CJ, Ribaudo HJ, Leon-Cruz J, Overton ET, Zanni MV, Malvestutto CD, Aberg JA, Kileel EM, Fitch KV, Van Schalkwyk M, Kumarasamy N, Martinez E, Santos BR, Joseph Y, Lo J, Siminski S, Melbourne K, Sponseller CA, Desvigne-Nickens P, Bloomfield GS, Currier JS, Hoffmann U, Douglas PS, Grinspoon SK; REPRIEVE Investigators. Patterns of Antiretroviral Therapy Use and Immunologic Profiles at Enrollment in the REPRIEVE Trial. J Infect Dis. 2020 Jul 9;222(Suppl 1):S8-S19. doi: 10.1093/infdis/jiaa259. PMID 32645162
- [Result] Smeaton LM, Kileel EM, Grinsztejn B, Gardner EM, Starr K, Murry ML, Desvigne-Nickens P, Alston-Smith B, Waclawiw MA, Cooper-Arnold K, Madruga JV, Sangle S, Fitch KV, Zanni MV, Douglas PS, Ribaudo HJ, Grinspoon SK, Klingman KL. Characteristics of REPRIEVE Trial Participants Identifying Across the Transgender Spectrum. J Infect Dis. 2020 Jul 9;222(Suppl 1):S31-S40. doi: 10.1093/infdis/jiaa213. PMID 32645160
- [Result] Zanni MV, Currier JS, Kantor A, Smeaton L, Rivard C, Taron J, Burdo TH, Badal-Faesen S, Lalloo UG, Pinto JA, Samaneka W, Valencia J, Klingman K, Allston-Smith B, Cooper-Arnold K, Desvigne-Nickens P, Lu MT, Fitch KV, Hoffman U, Grinspoon SK, Douglas PS, Looby SE. Correlates and Timing of Reproductive Aging Transitions in a Global Cohort of Midlife Women With Human Immunodeficiency Virus: Insights From the REPRIEVE Trial. J Infect Dis. 2020 Jul 9;222(Suppl 1):S20-S30. doi: 10.1093/infdis/jiaa214. PMID 32645159
- [Result] Neilan TG, Nguyen KL, Zaha VG, Chew KW, Morrison L, Ntusi NAB, Toribio M, Awadalla M, Drobni ZD, Nelson MD, Burdo TH, Van Schalkwyk M, Sax PE, Skiest DJ, Tashima K, Landovitz RJ, Daar E, Wurcel AG, Robbins GK, Bolan RK, Fitch KV, Currier JS, Bloomfield GS, Desvigne-Nickens P, Douglas PS, Hoffmann U, Grinspoon SK, Ribaudo H, Dawson R, Goetz MB, Jain MK, Warner A, Szczepaniak LS, Zanni MV. Myocardial Steatosis Among Antiretroviral Therapy-Treated People With Human Immunodeficiency Virus Participating in the REPRIEVE Trial. J Infect Dis. 2020 Jul 9;222(Suppl 1):S63-S69. doi: 10.1093/infdis/jiaa245. PMID 32645158
- [Result] Douglas PS, Umbleja T, Bloomfield GS, Fichtenbaum CJ, Zanni MV, Overton ET, Fitch KV, Kileel EM, Aberg JA, Currier J, Sponseller CA, Melbourne K, Avihingsanon A, Bustorff F, Estrada V, Ruxrungtham K, Saumoy M, Navar AM, Hoffmann U, Ribaudo HJ, Grinspoon S. Cardiovascular Risk and Health Among People With Human Immunodeficiency Virus (HIV) Eligible for Primary Prevention: Insights From the REPRIEVE Trial. Clin Infect Dis. 2021 Dec 6;73(11):2009-2022. doi: 10.1093/cid/ciab552. PMID 34134131
- [Result] Hoffmann U, Lu MT, Foldyna B, Zanni MV, Karady J, Taron J, Zhai BK, Burdo T, Fitch KV, Kileel EM, Williams K, Fichtenbaum CJ, Overton ET, Malvestutto C, Aberg J, Currier J, Sponseller CA, Melbourne K, Floris-Moore M, Van Dam C, Keefer MC, Koletar SL, Douglas PS, Ribaudo H, Mayrhofer T, Grinspoon SK; REPRIEVE trial. Assessment of Coronary Artery Disease With Computed Tomography Angiography and Inflammatory and Immune Activation Biomarkers Among Adults With HIV Eligible for Primary Cardiovascular Prevention. JAMA Netw Open. 2021 Jun 1;4(6):e2114923. doi: 10.1001/jamanetworkopen.2021.14923. PMID 34185068
- [Result] Kileel EM, Lo J, Malvestutto C, Fitch KV, Zanni MV, Fichtenbaum CJ, Overton ET, Okeke NL, Kumar P, Joao E, Aberg JA, Martinez E, Currier JS, Douglas PS, Ribaudo HJ, Grinspoon SK. Assessment of Obesity and Cardiometabolic Status by Integrase Inhibitor Use in REPRIEVE: A Propensity-Weighted Analysis of a Multinational Primary Cardiovascular Prevention Cohort of People With Human Immunodeficiency Virus. Open Forum Infect Dis. 2021 Nov 20;8(12):ofab537. doi: 10.1093/ofid/ofab537. eCollection 2021 Dec. PMID 34888395
- [Result] Fulda ES, Fitch KV, Overton ET, Zanni MV, Aberg JA, Currier JS, Lu MT, Malvestutto C, Fichtenbaum CJ, Martinez E, Umbleja T, Douglas PS, Ribaudo HJ, Grinspoon SK. COVID-19 Vaccination Rates in a Global HIV Cohort. J Infect Dis. 2022 Feb 15;225(4):603-607. doi: 10.1093/infdis/jiab575. PMID 34794178
- [Result] Bloomfield GS, Weir IR, Ribaudo HJ, Fitch KV, Fichtenbaum CJ, Moran LE, Bedimo R, de Filippi C, Morse CG, Piccini J, Zanni MV, Lu MT, Hoffmann U, Grinspoon SK, Douglas PS. Prevalence and Correlates of Electrocardiographic Abnormalities in Adults With HIV: Insights From the Randomized Trial to Prevent Vascular Events in HIV (REPRIEVE). J Acquir Immune Defic Syndr. 2022 Mar 1;89(3):349-359. doi: 10.1097/QAI.0000000000002877. PMID 35147583
- [Result] Erlandson KM, Fitch KV, McCallum SA, Ribaudo HJ, Overton ET, Zanni MV, Bloomfield GS, Brown TT, Fichtenbaum CJ, Bares S, Aberg JA, Douglas PS, Fulda ES, Santana-Bagur JL, Castro JG, Moran LE, Mave V, Supparatpinyo K, Ponatshego PL, Schechter M, Grinspoon SK. Geographical Differences in the Self-Reported Functional Impairment of People With Human Immunodeficiency Virus (HIV) and Associations With Cardiometabolic Risk. Clin Infect Dis. 2022 Sep 30;75(7):1154-1163. doi: 10.1093/cid/ciac098. PMID 35165682
- [Result] Looby SE, Kantor A, Burdo TH, Currier JS, Fichtenbaum CJ, Overton ET, Aberg JA, Malvestutto CD, Bloomfield GS, Erlandson KM, Cespedes M, Kallas EG, Masia M, Thornton AC, Smith MD, Flynn JM, Kileel EM, Fulda E, Fitch KV, Lu MT, Douglas PS, Grinspoon SK, Ribaudo HJ, Zanni MV. Factors Associated With Systemic Immune Activation Indices in a Global Primary Cardiovascular Disease Prevention Cohort of People With Human Immunodeficiency Virus on Antiretroviral Therapy. Clin Infect Dis. 2022 Oct 12;75(8):1324-1333. doi: 10.1093/cid/ciac166. PMID 35235653
- [Result] Overton ET, Weir IR, Zanni MV, Fischinger S, MacArthur RD, Aberg JA, Fitch KV, Frank M, Albrecht H, Goodenough E, Rhame FS, Fichtenbaum CJ, Bloomfield GS, Malvestutto C, Supparatpinyo K, McCallum S, Douglas PS, Alter G, Ribaudo H, Grinspoon SK. Asymptomatic SARS-CoV-2 Infection Is Common Among ART-Treated People With HIV. J Acquir Immune Defic Syndr. 2022 Aug 1;90(4):377-381. doi: 10.1097/QAI.0000000000003000. PMID 35413022
- [Result] Fitch KV, McCallum SA, Erlandson KM, Overton ET, Zanni MV, Fichtenbaum C, Aberg JA, Fulda ES, Kileel EM, Moran LE, Bloomfield GS, Novak RM, Perez-Frontera S, Abrams-Downey A, Pierone G Jr, Kumarasamy N, Ruxrungtham K, Mngqibisa R, Douglas PS, Ribaudo HJ, Grinspoon SK. Diet in a global cohort of adults with HIV at low-to-moderate traditional cardiovascular disease risk. AIDS. 2022 Nov 15;36(14):1997-2003. doi: 10.1097/QAD.0000000000003344. Epub 2022 Jul 27. PMID 35876637
- [Result] Kolossvary M, deFilippi C, Lu MT, Zanni MV, Fulda ES, Foldyna B, Ribaudo H, Mayrhofer T, Collier AC, Bloomfield GS, Fichtenbaum C, Overton ET, Aberg JA, Currier J, Fitch KV, Douglas PS, Grinspoon SK. Proteomic Signature of Subclinical Coronary Artery Disease in People With HIV: Analysis of the REPRIEVE Mechanistic Substudy. J Infect Dis. 2022 Nov 11;226(10):1809-1822. doi: 10.1093/infdis/jiac196. PMID 35535576
- [Result] Zanni MV, Foldyna B, McCallum S, Burdo TH, Looby SE, Fitch KV, Fulda ES, Autissier P, Bloomfield GS, Malvestutto CD, Fichtenbaum CJ, Overton ET, Aberg JA, Erlandson KM, Campbell TB, Ellsworth GB, Sheth AN, Taiwo B, Currier JS, Hoffmann U, Lu MT, Douglas PS, Ribaudo HJ, Grinspoon SK. Sex Differences in Subclinical Atherosclerosis and Systemic Immune Activation/Inflammation Among People With Human Immunodeficiency Virus in the United States. Clin Infect Dis. 2023 Jan 13;76(2):323-334. doi: 10.1093/cid/ciac767. PMID 36101518
- [Result] Schnittman SR, Lu MT, Mayrhofer T, Burdo TH, Fitch KV, McCallum S, Fulda ES, Zanni MV, Foldyna B, Malvestutto C, Fichtenbaum CJ, Aberg JA, Bloomfield GS, Overton ET, Currier J, Tebas P, Sha BE, Ribaudo HJ, Flynn JM, Douglas PS, Erlandson KM, Grinspoon SK. Cytomegalovirus Immunoglobulin G (IgG) Titer and Coronary Artery Disease in People With Human Immunodeficiency Virus (HIV). Clin Infect Dis. 2023 Feb 8;76(3):e613-e621. doi: 10.1093/cid/ciac662. PMID 35975297
- [Result] Douglas PS, McCallum S, Lu MT, Umbleja T, Fitch KV, Foldyna B, Zanni MV, Fulda ES, Bloomfield GS, Fichtenbaum CJ, Overton ET, Aberg JA, Malvestutto CD, Burdo TH, Arduino RC, Ho KS, Yin MT, Ribaudo HJ, Grinspoon SK. Ideal cardiovascular health, biomarkers, and coronary artery disease in persons with HIV. AIDS. 2023 Mar 1;37(3):423-434. doi: 10.1097/QAD.0000000000003418. Epub 2022 Nov 18. PMID 36525544
- [Result] Fulda ES, Fichtenbaum CJ, Kileel EM, Zanni MV, Aberg JA, Malvestutto C, Cardoso SW, Berzins B, Lira R, Harden R, Robbins G, Martinez M, Nieves SD, McCallum S, Cruz JL, Umbleja T, Sprenger H, Giguel F, Bone F, Wood K, Byroads M, Paradis K, Lu MT, Douglas PS, Ribaudo HJ, Grinspoon SK, Fitch KV; REPRIEVE Investigators. The importance of methods for site performance evaluation in REPRIEVE, a longitudinal, global, multicenter trial. Contemp Clin Trials. 2023 Jan;124:107035. doi: 10.1016/j.cct.2022.107035. Epub 2022 Nov 30. PMID 36462699
- [Result] Schnittman SR, Jung W, Fitch KV, Zanni MV, McCallum S, Lee JS, Shin S, Davis BJ, Fulda ES, Diggs MR, Giguel F, Chinchay R, Sheth AN, Fichtenbaum CJ, Malvestutto C, Aberg JA, Currier J, Lauffenburger DA, Douglas PS, Ribaudo HJ, Alter G, Grinspoon SK. Effect of host factors and COVID-19 infection on the humoral immune repertoire in treated HIV. JCI Insight. 2023 Mar 8;8(5):e166848. doi: 10.1172/jci.insight.166848. PMID 36805331
- [Result] Kileel EM, Malvestutto CD, Lo J, Fitch KV, Fichtenbaum CJ, Aberg JA, Zanni MV, Martinez E, Okeke NL, Kumar P, Joao E, Bares SH, Berrner D, Smieja M, Roa JC, McCallum S, Douglas PS, Ribaudo HJ, Grinspoon SK. Changes in Body Mass Index with Longer-term Integrase Inhibitor Use: A Longitudinal Analysis of Data from the Randomized Trial to Prevent Vascular Events in Human Immunodeficiency Virus (REPRIEVE). Clin Infect Dis. 2023 Jun 8;76(11):2010-2013. doi: 10.1093/cid/ciad107. PMID 36825498
- [Result] Schnittman SR, Kitch DW, Swartz TH, Burdo TH, Fitch KV, McCallum S, Flynn JM, Fulda ES, Diggs MR, Stapleton JT, Casado JL, Taron J, Currier JS, Zanni MV, Malvestutto C, Fichtenbaum CJ, Aberg JA, Ribaudo HJ, Lu MT, Douglas PS, Grinspoon SK. Coronary Artery Plaque Composition and Severity Relate to the Inflammasome in People With Treated Human Immunodeficiency Virus. Open Forum Infect Dis. 2023 Mar 1;10(3):ofad106. doi: 10.1093/ofid/ofad106. eCollection 2023 Mar. PMID 36998633
- [Result] Kolossvary M, deFilippi C, McCallum S, Fitch KV, Diggs MR, Fulda ES, Ribaudo HJ, Fichtenbaum CJ, Aberg JA, Malvestutto CD, Currier JS, Casado JL, Gutierrez F, Sereti I, Douglas PS, Zanni MV, Grinspoon SK. Identification of pre-infection markers and differential plasma protein expression following SARS-CoV-2 infection in people living with HIV. EBioMedicine. 2023 Apr;90:104538. doi: 10.1016/j.ebiom.2023.104538. Epub 2023 Mar 24. PMID 36966617
- [Result] Foldyna B, Mayrhofer T, Zanni MV, Lyass A, Barve R, Karady J, McCallum S, Burdo TH, Fitch KV, Paradis K, Fulda ES, Diggs MR, Bloomfield GS, Malvestutto CD, Fichtenbaum CJ, Aberg JA, Currier JS, Ribaudo HJ, Hoffmann U, Lu MT, Douglas PS, Grinspoon SK. Pericoronary Adipose Tissue Density, Inflammation, and Subclinical Coronary Artery Disease Among People With HIV in the REPRIEVE Cohort. Clin Infect Dis. 2023 Dec 15;77(12):1676-1686. doi: 10.1093/cid/ciad419. PMID 37439633
- [Result] Grinspoon SK, Fitch KV, Zanni MV, Fichtenbaum CJ, Umbleja T, Aberg JA, Overton ET, Malvestutto CD, Bloomfield GS, Currier JS, Martinez E, Roa JC, Diggs MR, Fulda ES, Paradis K, Wiviott SD, Foldyna B, Looby SE, Desvigne-Nickens P, Alston-Smith B, Leon-Cruz J, McCallum S, Hoffmann U, Lu MT, Ribaudo HJ, Douglas PS; REPRIEVE Investigators. Pitavastatin to Prevent Cardiovascular Disease in HIV Infection. N Engl J Med. 2023 Aug 24;389(8):687-699. doi: 10.1056/NEJMoa2304146. Epub 2023 Jul 23. PMID 37486775
- [Result] Lake JE, Taron J, Ribaudo HJ, Leon-Cruz J, Utay NS, Swaminathan S, Fitch KV, Kileel EM, Paradis K, Fulda ES, Ho KS, Luetkemeyer AF, Johnston CD, Zanni MV, Douglas PS, Grinspoon SK, Lu MT, Fichtenbaum CJ; REPRIEVE Trial Investigators. Hepatic steatosis and nonalcoholic fatty liver disease are common and associated with cardiometabolic risk in a primary prevention cohort of people with HIV. AIDS. 2023 Nov 15;37(14):2149-2159. doi: 10.1097/QAD.0000000000003671. Epub 2023 Jul 27. PMID 37503623
- [Result] Schnittman SR, Kolossvary M, Beck-Engeser G, Fitch KV, Ambayec GC, Nance RM, Zanni MV, Diggs M, Chan F, McCallum S, Toribio M, Bamford L, Fichtenbaum CJ, Eron JJ, Jacobson JM, Mayer KH, Malvestutto C, Bloomfield GS, Moore RD, Umbleja T, Saag MS, Aberg JA, Currier JS, Delaney JAC, Martin JN, Lu MT, Douglas PS, Ribaudo HJ, Crane HM, Hunt PW, Grinspoon SK. Biological and Clinical Implications of the Vascular Endothelial Growth Factor Coreceptor Neuropilin-1 in Human Immunodeficiency Virus. Open Forum Infect Dis. 2023 Sep 8;10(10):ofad467. doi: 10.1093/ofid/ofad467. eCollection 2023 Oct. PMID 37869406
- [Result] Bhattacharya R, Uddin MM, Patel AP, Niroula A, Finneran P, Bernardo R, Fitch KV, Lu MT, Bloomfield GS, Malvestutto C, Aberg JA, Fichtenbaum CJ, Hornsby W, Ribaudo HJ, Libby P, Ebert BL, Zanni MV, Douglas PS, Grinspoon SK, Natarajan P. Risk factors for clonal hematopoiesis of indeterminate potential in people with HIV: a report from the REPRIEVE trial. Blood Adv. 2024 Feb 27;8(4):959-967. doi: 10.1182/bloodadvances.2023011324. PMID 38197863
- [Result] Lu MT, Ribaudo H, Foldyna B, Zanni MV, Mayrhofer T, Karady J, Taron J, Fitch KV, McCallum S, Burdo TH, Paradis K, Hedgire SS, Meyersohn NM, DeFilippi C, Malvestutto CD, Sturniolo A, Diggs M, Siminski S, Bloomfield GS, Alston-Smith B, Desvigne-Nickens P, Overton ET, Currier JS, Aberg JA, Fichtenbaum CJ, Hoffmann U, Douglas PS, Grinspoon SK; REPRIEVE Trial Writing Group. Effects of Pitavastatin on Coronary Artery Disease and Inflammatory Biomarkers in HIV: Mechanistic Substudy of the REPRIEVE Randomized Clinical Trial. JAMA Cardiol. 2024 Apr 1;9(4):323-334. doi: 10.1001/jamacardio.2023.5661. PMID 38381407
- [Result] Zou RS, Ruan Y, Truong B, Bhattacharya R, Lu MT, Karady J, Bernardo R, Finneran P, Hornsby W, Fitch KV, Ribaudo HJ, Zanni MV, Douglas PS, Grinspoon SK, Patel AP, Natarajan P. Polygenic Scores and Preclinical Cardiovascular Disease in Individuals With HIV: Insights From the REPRIEVE Trial. J Am Heart Assoc. 2024 Apr 2;13(7):e033413. doi: 10.1161/JAHA.123.033413. Epub 2024 Mar 27. PMID 38533953
- [Result] Grinspoon SK, Ribaudo HJ, Douglas PS. Trial Update of Pitavastatin to Prevent Cardiovascular Events in HIV Infection. N Engl J Med. 2024 May 2;390(17):1626-1628. doi: 10.1056/NEJMc2400870. No abstract available. PMID 38692296
- [Derived] Foldyna B, Hadzic I, Mayrhofer T, Karady J, Taron J, Kolossvary M, Raghu VK, McCallum S, Paradis K, Diggs MR, Chu SM, Lu AB, Somboonwit C, Bernardino JI, Dube MP, Sponseller CA, Zanni MV, Bloomfield GS, Malvestutto CD, Fichtenbaum CJ, Aberg JA, Currier JS, Ribaudo HJ, Douglas PS, Lu MT, Grinspoon SK. Statin Effects on Pericoronary Adipose Tissue Density in People With HIV: Insights From the REPRIEVE Trial. JACC Cardiovasc Imaging. 2025 Nov 24:S1936-878X(25)00594-7. doi: 10.1016/j.jcmg.2025.10.012. Online ahead of print. PMID 41324519
- [Derived] Diggs MR, Chu SM, Fitch KV, Olefsky M, Watanabe MG, Erlandson KM, Lu AB, Bloomfield GS, Currier JS, Curran A, Eckard AR, Smith GHR, Sponseller CA, Fichtenbaum CJ, Malvestutto CD, Aberg JA, Foldyna B, Taron J, Karady J, Zanni MV, Douglas PS, Ribaudo HJ, Lu MT, Grinspoon SK. Health-related quality of life among people with HIV at low-to-moderate risk for atherosclerotic cardiovascular disease in the REPRIEVE Trial. AIDS. 2025 Nov 10. doi: 10.1097/QAD.0000000000004401. Online ahead of print. PMID 41217428
- [Derived] Xue L, Bhattacharya R, Uddin MM, Nakao T, Zou R, Patel A, Haidermota S, Niroula A, Viscosi V, Postupaka D, Bhatnagar A, Finneran P, Bernardo R, Diggs MR, Fitch KV, Chu SM, McCallum S, Currier JS, Fichtenbaum CJ, Malvestutto CD, Aberg JA, Bloomfield GS, Ribaudo HJ, Zanni MV, Libby P, Hornsby W, Lu MT, Douglas PS, Grinspoon SK, Natarajan P. Clonal Hematopoiesis and Major Adverse Cardiac Events in People With HIV: Insights From the REPRIEVE Trial. Arterioscler Thromb Vasc Biol. 2026 Jan;46(1):168-177. doi: 10.1161/ATVBAHA.125.322896. Epub 2025 Nov 6. PMID 41195533
- [Derived] Grinspoon SK, Zhao S, Martinez E, Fichtenbaum CJ, Chu SM, Diggs MR, Umbleja T, McCallum S, Fitch KV, Triant VA, Currier JS, Aberg JA, Malvestutto CD, Erlandson KM, Bloomfield GS, Lu MT, Douglas PS, Ribaudo HJ, Zanni MV. Risk Assessment in a Global CVD Prevention Cohort of People with HIV by PCE, PREVENT, and SCORE2. Clin Infect Dis. 2025 Sep 26:ciaf542. doi: 10.1093/cid/ciaf542. Online ahead of print. PMID 41004413
- [Derived] Kolossvary M, Sereti I, Zanni MV, Fichtenbaum CJ, Aberg JA, Bloomfield GS, Malvestutto CD, Currier JS, Chu SM, Diggs MR, Lu AB, deFilippi C, Foldyna B, McCallum S, Sponseller CA, Lu MT, Douglas PS, Ribaudo HJ, Grinspoon SK. Statin-dependent and -independent pathways are associated with major adverse cardiovascular events in people with HIV. J Clin Invest. 2025 Sep 9;135(22):e196021. doi: 10.1172/JCI196021. eCollection 2025 Nov 17. PMID 40924496
- [Derived] Davies Smith E, Douglas PS, McCallum S, Troendle J, Diggs MR, Lu AB, Chu SM, Umbleja T, Lu MT, Zanni MV, Grinspoon SK, Ribaudo HJ. Win Ratio Aligns With and Enhances Interpretation of REPRIEVE's Primary Findings. Clin Infect Dis. 2026 Feb 9;82(1):e89-e92. doi: 10.1093/cid/ciaf477. PMID 40888096
- [Derived] Corley MJ, Watanabe M, Pang APS, Dwaraka VB, Smith R, Samaneka W, Henn S, Munsiff S, Saumoy M, McCallum S, Fitch KV, Chu SM, Diggs MR, Aberg JA, Malvestutto CD, Fichtenbaum CJ, Currier JS, Zanni MV, Douglas PS, Lu MT, Landay AL, Erlandson KM, Ribaudo HJ, Grinspoon SK. Effect of Pitavastatin on Epigenetic Aging Biomarkers in People With HIV: Pilot Substudy of the REPRIEVE Trial. Clin Infect Dis. 2025 Jun 18:ciaf247. doi: 10.1093/cid/ciaf247. Online ahead of print. PMID 40576558
- [Derived] Fichtenbaum CJ, Malvestutto CD, Watanabe MG, Davies Smith E, Ribaudo HJ, McCallum S, Fitch KV, Currier JS, Diggs MR, Chu SM, Aberg JA, Lu MT, Valencia J, Gomez-Ayerbe C, Brar I, Valdez Madruga J, Bloomfield GS, Douglas PS, Zanni MV, Grinspoon SK; REPRIEVE Investigators. Effects of antiretrovirals on major adverse cardiovascular events in the REPRIEVE trial: a longitudinal cohort analysis. Lancet HIV. 2025 Jul;12(7):e496-e505. doi: 10.1016/S2352-3018(25)00043-8. Epub 2025 Jun 4. PMID 40482662
- [Derived] Lu MT, Ribaudo HJ, McCallum S, Zanni MV, deFilippi C, Taron J, Karady J, Foldyna B, Paradis K, Chu SM, Diggs MR, Burdo TH, Currier JS, Bloomfield GS, Fichtenbaum CJ, Malvestutto CD, Aberg JA, Mayrhofer T, Douglas PS, Grinspoon SK; REPRIEVE Investigators. Coronary Plaque, Inflammation, Subclinical Myocardial Injury, and Major Adverse Cardiovascular Events in the REPRIEVE Substudy. JACC Adv. 2025 Jun;4(6 Pt 1):101781. doi: 10.1016/j.jacadv.2025.101781. Epub 2025 May 14. PMID 40373520
- [Derived] Grinspoon SK, Watanabe M, Ribaudo HJ, Bloomfield GS, Fichtenbaum CJ, Umbleja T, Chu SM, Fitch KV, Diggs MR, Zhao S, Looby SE, Currier JS, Aberg JA, Malvestutto CD, Erlandson KM, Martinez E, Asupoto O, Gupta SK, Lopez-Bernaldo de Quiros JC, Nixon D, Bedimo R, Lu MT, Douglas PS, Zanni MV. Factors Affecting Risk of Cardiovascular Disease (CVD) Events in a Global CVD Prevention Cohort of People With HIV. Clin Infect Dis. 2026 Feb 4;81(6):e548-e557. doi: 10.1093/cid/ciaf210. PMID 40281648
- [Derived] Davies Smith E, Malvestutto C, Ribaudo HJ, Fichtenbaum CJ, Aberg JA, Watanabe M, Bloomfield GS, Currier JS, Chu SM, Fitch KV, Diggs MR, Bedimo R, Valencia J, Gomez-Ayerbe C, Brar I, Madruga JV, Lu MT, Douglas PS, Zanni MV, Grinspoon SK. Cardiovascular Hazards of Abacavir- Versus Tenofovir-Containing Antiretroviral Therapies: Insights From an Analysis of the REPRIEVE Trial Cohort. Open Forum Infect Dis. 2025 Mar 21;12(4):ofaf177. doi: 10.1093/ofid/ofaf177. eCollection 2025 Apr. PMID 40207047
- [Derived] Diggs MR, Umbleja T, McCallum S, Zanni MV, Chu SM, Fitch KV, Bloomfield GS, Currier JS, Martinez E, Castle PE, Awwad A, Jain MK, Bedimo R, Hendricks B, Narrea J, Estrada V, Pinto J, Aberg JA, Malvestutto CD, Fichtenbaum CJ, Lu MT, Ribaudo HJ, Douglas PS, Grinspoon SK. Statin effects on the incidence of major non-cardiovascular disease events among a global cohort of people with HIV: a randomised controlled trial. Lancet HIV. 2025 Apr;12(4):e261-e272. doi: 10.1016/S2352-3018(24)00345-X. PMID 40180472
- [Derived] Grinspoon SK, Zanni MV, Triant VA, Kantor A, Umbleja T, Diggs MR, Chu SM, Fitch KV, Currier JS, Bloomfield GS, Casado JL, de la Pena M, Fantry LE, Gardner E, Aberg JA, Malvestutto CD, Fichtenbaum CJ, Lu MT, Ribaudo HJ, Douglas PS. Performance of the pooled cohort equations and D:A:D risk scores among individuals with HIV in a global cardiovascular disease prevention trial: a cohort study leveraging data from REPRIEVE. Lancet HIV. 2025 Feb;12(2):e118-e129. doi: 10.1016/S2352-3018(24)00276-5. Epub 2025 Jan 17. PMID 39832519
- [Derived] Kolossvary M, Schnittman SR, Zanni MV, Fitch KV, Fichtenbaum CJ, Aberg JA, Bloomfield GS, Malvestutto CD, Currier J, Diggs MR, deFilippi C, Eckard AR, Curran A, Centinbas M, Sadreyev R, Foldyna B, Mayrhofer T, Karady J, Taron J, McCallum S, Lu MT, Ribaudo HJ, Douglas PS, Grinspoon SK. Pitavastatin, Procollagen Pathways, and Plaque Stabilization in Patients With HIV: A Secondary Analysis of the REPRIEVE Randomized Clinical Trial. JAMA Cardiol. 2025 Mar 1;10(3):254-264. doi: 10.1001/jamacardio.2024.4115. PMID 39661372
- [Derived] Zanni MV, Umbleja T, Fichtenbaum CJ, Fitch KV, McCallum S, Aberg JA, Overton ET, Malvestutto CD, Bloomfield GS, Currier JS, Schnittman SR, Erlandson KM, Diggs MR, Foldyna B, Martinez E, Somboonwit C, Wang GP, Mushatt D, Connick E, Lu MT, Douglas PS, Ribaudo HJ, Grinspoon SK. Effects of Pitavastatin on COVID-19 Incidence and Seriousness Among a Global Cohort of People With HIV. Open Forum Infect Dis. 2024 Oct 10;11(10):ofae574. doi: 10.1093/ofid/ofae574. eCollection 2024 Oct. PMID 39435321
- [Derived] Fitch KV, Zanni MV, Manne-Goehler J, Diggs MR, Gattu AK, Currier JS, Bloomfield GS, Hsiao CB, Gupta SK, Aberg JA, Malvestutto CD, Fichtenbaum CJ, Lu MT, Douglas PS, Ribaudo HJ, Grinspoon SK. Diabetes Risk Factors in People With HIV Receiving Pitavastatin Versus Placebo for Cardiovascular Disease Prevention : A Randomized Trial. Ann Intern Med. 2024 Nov;177(11):1449-1461. doi: 10.7326/ANNALS-24-00944. Epub 2024 Oct 8. PMID 39374532
- [Derived] deFilippi C, McCallum S, Zanni MV, Fitch KV, Diggs MR, Bloomfield GS, Fichtenbaum CJ, Aberg JA, Malvestutto CD, Pinto-Martinez A, Stapleton A, Duggan J, Robbins GK, Taron J, Karady J, Foldyna B, Lu MT, Ribaudo HJ, Douglas PS, Grinspoon SK. Association of Cardiac Troponin T With Coronary Atherosclerosis in Asymptomatic Primary Prevention People With HIV. JACC Adv. 2024 Aug 16;3(9):101206. doi: 10.1016/j.jacadv.2024.101206. eCollection 2024 Sep. PMID 39253712
- [Derived] Erlandson KM, Umbleja T, Ribaudo HJ, Schrack JA, Overton ET, Fichtenbaum CJ, Fitch KV, Roa JC, Diggs MR, Wood K, Zanni MV, Bloomfield GS, Malvestutto C, Aberg JA, Rodriguez-Barradas MC, Morones RG, Breaux K, Douglas PS, Grinspoon SK, Brown TT. Pitavastatin Is Well-Tolerated With no Detrimental Effects on Physical Function. Clin Infect Dis. 2025 Feb 24;80(2):425-433. doi: 10.1093/cid/ciae422. PMID 39159048
- [Derived] Abidi MZ, Umbleja T, Overton ET, Burdo T, Flynn JM, Lu MT, Taron J, Schnittman SR, Fitch KV, Zanni MV, Fichtenbaum CJ, Malvestutto C, Aberg JA, Fulda ES, Eckard AR, Manne-Goehler J, Tuan JJ, Ribaudo HJ, Douglas PS, Grinspoon SK, Brown TT, Erlandson KM. Cytomegalovirus IgG is Associated With Physical Function But Not Muscle Density in People With HIV. J Acquir Immune Defic Syndr. 2024 Apr 15;95(5):470-478. doi: 10.1097/QAI.0000000000003377. PMID 38180893
- [Derived] Erlandson KM, Umbleja T, Lu MT, Taron J, Ribaudo HJ, Overton ET, Presti RM, Haas DW, Sax PE, Yin MT, Zhai BK, Louis R, Upadhyay N, Eslami P, Douglas PS, Zanni MV, Fitch KV, Fulda ES, Fichtenbaum CJ, Malvestutto CD, Grinspoon SK, Brown TT. Associations of Muscle Density and Area With Coronary Artery Plaque and Physical Function. J Acquir Immune Defic Syndr. 2023 Oct 1;94(2):174-184. doi: 10.1097/QAI.0000000000003244. PMID 37368931
- [Derived] Umbleja T, Brown TT, Overton ET, Ribaudo HJ, Schrack JA, Fitch KV, Douglas PS, Grinspoon SK, Henn S, Arduino RC, Rodriguez B, Benson CA, Erlandson KM. Physical Function Impairment and Frailty in Middle-Aged People Living With Human Immunodeficiency Virus in the REPRIEVE Trial Ancillary Study PREPARE. J Infect Dis. 2020 Jul 9;222(Suppl 1):S52-S62. doi: 10.1093/infdis/jiaa249. PMID 32645163
- See also: REPRIEVE Trial Website — http://reprievetrial.org/
- See also: Division of AIDS Table for Grading the Severity of Adult and Pediatric Adverse Events (DAIDS AE Grading Table), corrected Version 2.1, July 2017 — https://rsc.niaid.nih.gov/sites/default/files/daids-ae-grading-table-v2-nov2014.pdf
- See also: Clinical Safety Data Management: Definitions and Standards for Expedited Reporting E2A — https://database.ich.org/sites/default/files/E2A_Guideline.pdf

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled from March 26, 2015 to July 31, 2019.
Pre-assignment Details: 4 inadvertent duplicate enrollments of the same person were excluded. The total enrollment number of 7769 represents unique participants enrolled.
Period: Overall Study
Arm/Group | Pitavastatin | Placebo
Started | 3888 | 3881
Enrolled in Mechanistic Substudy | 402 | 402
Completed Mechanistic Substudy | 349 | 350
Completed | 3201 | 3201
Not Completed | 687 | 680
Not completed — Withdrawal by Subject | 315 | 324
Not completed — Lost to Follow-up | 258 | 249
Not completed — Unable to get to clinic | 69 | 60
Not completed — Physician Decision | 25 | 25
Not completed — Site Closure | 15 | 19
Not completed — Other | 5 | 3

BASELINE CHARACTERISTICS:
Population: All participants enrolled.
Groups:
- Total: Total of all reporting groups
Arm/Group | Pitavastatin | Placebo | Total
Number analyzed (Participants) | 3888 | 3881 | 7769
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 50 [45 to 55] | 50 [45 to 55] | 50 [45 to 55]
Age, Customized [Count of Participants; unit: Participants]
  40-49 years | 1842 | 1888 | 3730
  50-59 years | 1712 | 1649 | 3361
  ≥60 years | 334 | 344 | 678
Sex/Gender, Customized [Count of Participants; unit: Participants] — Gender identity was reported by the participants.
  Participants
    Cisgender | 3691 | 3683 | 7374
    Transgender | 63 | 64 | 127
    Not reported | 134 | 134 | 268
Sex: Female, Male [Count of Participants; unit: Participants] — Sex assigned at birth.
  Participants
    Female | 1211 | 1208 | 2419
    Male | 2677 | 2673 | 5350
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Ethnicity was reported by the participants according to the National Institutes of Health definition for participants in the United States (including Puerto Rico) and Canada. "Unknown or Not Reported" include participants who reported that their ethnicity is unknown or that they do not wish to report their ethnicity. Population: Participants in the United States (including Puerto Rico) and Canada. Because the ethnicity definition is not applicable to other geographic regions, they were excluded from the measure analysis population.
  Participants
    number analyzed (Participants) | 1957 | 1961 | 3918
    Hispanic or Latino | 366 | 332 | 698
    Not Hispanic or Latino | 1575 | 1611 | 3186
    Unknown or Not Reported | 16 | 18 | 34
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Race was reported by the participants. "Other" race includes participants who identified as native or indigenous to the enrollment region, as having more than one race, or as having an unknown race.
  Participants
    Black | 1569 | 1639 | 3208
    White | 1364 | 1340 | 2704
    Asian | 571 | 567 | 1138
    Other | 384 | 335 | 719
Region of Enrollment [Number; unit: participants]
  Haiti | 69 | 71 | 140
  United States | 1897 | 1890 | 3787
  Thailand | 304 | 286 | 590
  India | 246 | 258 | 504
  Spain | 106 | 107 | 213
  Canada | 60 | 71 | 131
  Botswana | 145 | 136 | 281
  Brazil | 546 | 553 | 1099
  South Africa | 282 | 288 | 570
  Uganda | 96 | 85 | 181
  Zimbabwe | 62 | 63 | 125
  Peru | 75 | 73 | 148
Global burden of disease (GBD) region [Count of Participants; unit: Participants]
  High income | 2044 | 2051 | 4095
  Latin America and Caribbean | 709 | 714 | 1423
  Southeast or East Asia | 304 | 286 | 590
  South Asia | 246 | 258 | 504
  Sub-Saharan Africa | 585 | 572 | 1157
Atherosclerotic Cardiovascular Disease (ASCVD) risk score [Count of Participants; unit: Participants] — 10-Year Atherosclerotic Cardiovascular Disease (ASCVD) risk score is calculated based on age, sex, race, systolic blood pressure, total and high-density lipoprotein cholesterol, hypertension treatment, smoking history and presence of diabetes. It is measured on a continuous scale, with 0-<5% considered low risk, 5-<7.5% borderline risk, 7.5-<20% intermediate risk, and ≥20% high risk according to the American College of Cardiology and American Heart Association. More granular categories were used to describe REPRIEVE participants, given the eligibility criterion of low to moderate CVD risk.
  Participants
    0 - <2.5% | 1096 | 1060 | 2156
    2.5 - <5% | 1030 | 1025 | 2055
    5 - <7.5% | 934 | 960 | 1894
    7.5 - 10% | 540 | 561 | 1101
    ≥10% | 288 | 275 | 563
Nadir CD4 cell count [Count of Participants; unit: Participants]
  <200 cells/mm^3 | 1890 | 1911 | 3801
  200 - 349 cells/mm^3 | 1019 | 1022 | 2041
  ≥350 cells/mm^3 | 839 | 825 | 1664
  Unknown | 140 | 123 | 263
CD4 cell count [Count of Participants; unit: Participants]
  ≤500 cells/mm^3 | 1257 | 1253 | 2510
  >500 cells/mm^3 | 2631 | 2628 | 5259
HIV-1 RNA [Count of Participants; unit: Participants] — The assays that were used for testing varied, including assays with a lower limit of quantification (LLQ) of 20 to 400 copies/mL. Population: The level of HIV-1 RNA was collected if data were available through standard care.
  Participants
    number analyzed (Participants) | 3009 | 2988 | 5997
    <LLQ | 2641 | 2609 | 5250
    LLQ - <400 copies/mL | 305 | 312 | 617
    ≥400 copies/mL | 63 | 67 | 130
Pre-existing diabetes [Count of Participants; unit: Participants] | 24 | 14 | 38
Mechanistic Substudy: Presence of Non-calcified Plaque (NCP) [Count of Participants; unit: Participants] — Presence of NCP defined as evidence of NCP based on the qualitative read of the CT scan. Note that presence of NCP based on the qualitative read does not necessarily mean that NCP volume can be quantified based on the quantitative read or vice versa. Population: Participants enrolled in the Mechanistic Substudy with paired CT scans (entry and year 2) and data on this measure available.
  Participants
    number analyzed (Participants) | 321 | 323 | 644
    NCP present | 132 | 139 | 271
    NCP not present | 189 | 184 | 373
Mechanistic Substudy: NCP Volume [Mean (Standard Deviation); unit: mm^3] — NCP was defined as plaque voxels with attenuation <350 Hounsfield Units (HU) based on the quantitative read of the CT scan. If no quantitative result was available, structural zeroes were assigned if no NCP was present based on the qualitative read. Population: Participants enrolled in the Mechanistic Substudy with paired CT scans (entry and year 2) and data on this measure available.
  mm^3
    number analyzed (Participants) | 290 | 297 | 587
    (all) | 52.3 (193.5) | 57.7 (109.2) | 55.1 (156.5)
Mechanistic Substudy: Total Plaque Volume [Mean (Standard Deviation); unit: mm^3] — Population: Participants enrolled in the Mechanistic Substudy with paired CT scans (entry and year 2) and data on this measure available.
  mm^3
    number analyzed (Participants) | 302 | 309 | 611
    (all) | 65.6 (211.7) | 72.2 (135.9) | 69.0 (176.8)

OUTCOME MEASURES:

1. Primary Outcome: Incidence Rate of Major Adverse Cardiovascular Event (MACE)
Description: MACE is a composite of cardiovascular (CV) death, myocardial infarction, hospitalization for unstable angina, stroke, transient ischemic attack (TIA), peripheral arterial ischemia, coronary, carotid or peripheral arterial revascularization, or death from an undetermined cause. The incidence rates were estimated based on time to the first event using Poisson distribution, with follow-up time censored at last contact. The treatment effect was estimated via cause-specific relative hazard (i.e. hazard ratio) of prescribed pitavastatin compared to placebo from Cox proportional hazards models, stratified by screening CD4 count and sex. Non-CV deaths (without preceding event of interest) were treated as competing events and censored. Treatment discontinuation was ignored, including the initiation of statin therapy as part of clinical care (intention to treat policy).
Time Frame: From entry through end of study. Follow-up time varied depending on time of enrollment (the median follow-up time was 5.6 years).
Population: All participants enrolled according to the randomized treatment group.
Measure: Number (95% Confidence Interval); unit: events per 1000 person-years
Arm/Group | Pitavastatin | Placebo
Number analyzed (Participants) | 3888 | 3881
events per 1000 person-years | 4.95 [4.07 to 6.03] | 7.77 [6.64 to 9.08]
Statistical Analysis 1: Comparison: Pitavastatin vs Placebo; Test type: Superiority; Hazard Ratio (HR) = 0.64, 95% CI 2-sided [0.48 to 0.84] — Hazard ratio is shown as pitavastatin/placebo. Two-sided 95% repeated confidence interval that adjusts for interim looks according to the realized Lan and DeMets implementation of the O'Brien-Fleming sequential stopping boundary is presented

2. Secondary Outcome: Incidence Rate of Cardiac Ischemia or Myocardial Infarction
Description: Cardiac ischemia or myocardial infarction component of the primary composite MACE outcome. The incidence rates were estimated based on time to the first event using Poisson distribution, with follow-up time censored at last contact. The treatment effect was estimated via cause-specific relative hazard (i.e. hazard ratio) of prescribed pitavastatin compared to placebo from Cox proportional hazards models, stratified by screening CD4 count and sex. Deaths (without preceding event of interest) were treated as competing events and censored. Treatment discontinuation was ignored, including the initiation of statin therapy as part of clinical care (intention to treat policy).
Time Frame: as for outcome 1
Population: All participants enrolled according to the randomized treatment group.
Measure: Number (95% Confidence Interval); unit: events per 1000 person-years
Arm/Group | Pitavastatin | Placebo
Number analyzed (Participants) | 3888 | 3881
events per 1000 person-years | 1.48 [1.03 to 2.11] | 2.65 [2.03 to 3.46]
Statistical Analysis 1: Comparison: Pitavastatin vs Placebo; Test type: Superiority; Hazard Ratio (HR) = 0.56, 95% CI 2-sided [0.36 to 0.87] — Hazard ratio is shown as pitavastatin/placebo

3. Secondary Outcome: Incidence Rate of Cerebrovascular Event (Stroke or TIA)
Description: Cerebrovascular event (stroke or TIA) component of the primary composite MACE outcome. The incidence rates were estimated based on time to the first event using Poisson distribution, with follow-up time censored at last contact. The treatment effect was estimated via cause-specific relative hazard (i.e. hazard ratio) of prescribed pitavastatin compared to placebo from Cox proportional hazards models, stratified by screening CD4 count and sex. Deaths (without preceding event of interest) were treated as competing events and censored. Treatment discontinuation was ignored, including the initiation of statin therapy as part of clinical care (intention to treat policy).
Time Frame: as for outcome 1
Population: All participants enrolled according to the randomized treatment group.
Measure: Number (95% Confidence Interval); unit: events per 1000 person-years
Arm/Group | Pitavastatin | Placebo
Number analyzed (Participants) | 3888 | 3881
events per 1000 person-years | 1.53 [1.07 to 2.17] | 2.46 [1.86 to 3.24]
Statistical Analysis 1: Comparison: Pitavastatin vs Placebo; Test type: Superiority; Hazard Ratio (HR) = 0.62, 95% CI 2-sided [0.40 to 0.97] — Hazard ratio is shown as pitavastatin/placebo

4. Secondary Outcome: Incidence Rate of Peripheral Arterial Ischemia
Description: Peripheral arterial ischemia component of the primary composite MACE outcome. The incidence rates were estimated based on time to the first event using Poisson distribution, with follow-up time censored at last contact. The treatment effect was estimated via cause-specific relative hazard (i.e. hazard ratio) of prescribed pitavastatin compared to placebo from Cox proportional hazards models, stratified by screening CD4 count and sex. Deaths (without preceding event of interest) were treated as competing events and censored. Treatment discontinuation was ignored, including the initiation of statin therapy as part of clinical care (intention to treat policy).
Time Frame: as for outcome 1
Population: All participants enrolled according to the randomized treatment group.
Measure: Number (95% Confidence Interval); unit: events per 1000 person-years
Arm/Group | Pitavastatin | Placebo
Number analyzed (Participants) | 3888 | 3881
events per 1000 person-years | 0.10 [0.02 to 0.39] | 0.15 [0.05 to 0.45]
Statistical Analysis 1: Comparison: Pitavastatin vs Placebo; Test type: Superiority; Hazard Ratio (HR) = 0.67, 95% CI 2-sided [0.11 to 4.02] — Hazard ratio is shown as pitavastatin/placebo

5. Secondary Outcome: Incidence Rate of Death From CV Causes
Description: CV death component of the primary composite MACE outcome. The incidence rates were estimated based on time to the first event using Poisson distribution, with follow-up time censored at last contact. The treatment effect was estimated via cause-specific relative hazard (i.e. hazard ratio) of prescribed pitavastatin compared to placebo from Cox proportional hazards models, stratified by screening CD4 count and sex. Non-CV deaths and deaths from undetermined causes were treated as competing events and censored. Treatment discontinuation was ignored, including the initiation of statin therapy as part of clinical care (intention to treat policy).
Time Frame: as for outcome 1
Population: All participants enrolled according to the randomized treatment group.
Measure: Number (95% Confidence Interval); unit: events per 1000 person-years
Arm/Group | Pitavastatin | Placebo
Number analyzed (Participants) | 3888 | 3881
events per 1000 person-years | 0.69 [0.41 to 1.16] | 0.98 [0.63 to 1.51]
Statistical Analysis 1: Comparison: Pitavastatin vs Placebo; Test type: Superiority; Hazard Ratio (HR) = 0.70, 95% CI 2-sided [0.35 to 1.38] — Hazard ratio is shown as pitavastatin/placebo

6. Secondary Outcome: Incidence Rate of Death From CV or Undetermined Causes
Description: CV or undetermined death component of the primary composite MACE outcome. The incidence rates were estimated based on time to the first event using Poisson distribution, with follow-up time censored at last contact. The treatment effect was estimated via cause-specific relative hazard (i.e. hazard ratio) of prescribed pitavastatin compared to placebo from Cox proportional hazards models, stratified by screening CD4 count and sex. Non-CV deaths were treated as competing events and censored. Treatment discontinuation was ignored, including the initiation of statin therapy as part of clinical care (intention to treat policy).
Time Frame: as for outcome 1
Population: All participants enrolled according to the randomized treatment group.
Measure: Number (95% Confidence Interval); unit: events per 1000 person-years
Arm/Group | Pitavastatin | Placebo
Number analyzed (Participants) | 3888 | 3881
events per 1000 person-years | 1.72 [1.23 to 2.39] | 2.54 [1.94 to 3.33]
Statistical Analysis 1: Comparison: Pitavastatin vs Placebo; Test type: Superiority; Hazard Ratio (HR) = 0.67, 95% CI 2-sided [0.44 to 1.03] — Hazard ratio is shown as pitavastatin/placebo

7. Secondary Outcome: Incidence Rate of Cardiac Catheterization or Revascularization
Description: Cardiac cardiac catheterization or revascularization component of the primary composite MACE outcome. The incidence rates were estimated based on time to the first event using Poisson distribution, with follow-up time censored at last contact. The treatment effect was estimated via cause-specific relative hazard (i.e. hazard ratio) of prescribed pitavastatin compared to placebo from Cox proportional hazards models, stratified by screening CD4 count and sex. Deaths (without preceding event of interest) were treated as competing events and censored. Treatment discontinuation was ignored, including the initiation of statin therapy as part of clinical care (intention to treat policy).
Time Frame: as for outcome 1
Population: All participants enrolled according to the randomized treatment group.
Measure: Number (95% Confidence Interval); unit: events per 1000 person-years
Arm/Group | Pitavastatin | Placebo
Number analyzed (Participants) | 3888 | 3881
events per 1000 person-years | 1.08 [0.71 to 1.64] | 1.77 [1.27 to 2.45]
Statistical Analysis 1: Comparison: Pitavastatin vs Placebo; Test type: Superiority; Hazard Ratio (HR) = 0.62, 95% CI 2-sided [0.36 to 1.05]; Hazard ratio is shown as pitavastatin/placebo

8. Secondary Outcome: Incidence Rate of Carotid or Cerebrovascular Revascularization
Description: Carotid or cerebrovascular revascularization component of the primary composite MACE outcome. The incidence rates were estimated based on time to the first event using Poisson distribution, with follow-up time censored at last contact. The treatment effect was estimated via cause-specific relative hazard (i.e. hazard ratio) of prescribed pitavastatin compared to placebo from Cox proportional hazards models, stratified by screening CD4 count and sex. Deaths (without preceding event of interest) were treated as competing events and censored. Treatment discontinuation was ignored, including the initiation of statin therapy as part of clinical care (intention to treat policy).
Time Frame: as for outcome 1
Population: All participants enrolled according to the randomized treatment group.
Measure: Number (95% Confidence Interval); unit: events per 1000 person-years
Arm/Group | Pitavastatin | Placebo
Number analyzed (Participants) | 3888 | 3881
events per 1000 person-years | 0 [NA to NA] — No events were observed in the pitavastatin group. Confidence interval could not be estimated. | 0 [NA to NA] — No events were observed in the placebo group. Confidence interval could not be estimated.

9. Secondary Outcome: Incidence Rate of Peripheral Arterial Revascularization
Description: Peripheral arterial revascularization component of the primary composite MACE outcome. The incidence rates were estimated based on time to the first event using Poisson distribution, with follow-up time censored at last contact. The treatment effect was estimated via cause-specific relative hazard (i.e. hazard ratio) of prescribed pitavastatin compared to placebo from Cox proportional hazards models, stratified by screening CD4 count and sex. Deaths (without preceding event of interest) were treated as competing events and censored. Treatment discontinuation was ignored, including the initiation of statin therapy as part of clinical care (intention to treat policy).
Time Frame: as for outcome 1
Population: All participants enrolled according to the randomized treatment group.
Measure: Number (95% Confidence Interval); unit: events per 1000 person-years
Arm/Group | Pitavastatin | Placebo
Number analyzed (Participants) | 3888 | 3881
events per 1000 person-years | 0 [NA to NA] — No events were observed in the pitavastatin group. Confidence interval could not be estimated. | 0.29 [0.13 to 0.65]
Statistical Analysis 1: Comparison: Pitavastatin vs Placebo; Test type: Superiority; Hazard Ratio (HR) = 0.00, 95% CI 2-sided [0.00 to 0.54]; Hazard ratio is shown as pitavastatin/placebo. Estimation of the confidence interval used a Bayes analysis with a non-informative prior using adaptive rejection Metropolis sampling. In this case, the interval shown is a 95% highest posterior density (HPD) interval

10. Secondary Outcome: Incidence Rate of MACE or Death
Description: A composite outcome including MACE and death from any cause. The incidence rates were estimated based on time to the first event using Poisson distribution, with follow-up time censored at last contact. The treatment effect was estimated via relative hazard (i.e. hazard ratio) of prescribed pitavastatin compared to placebo from Cox proportional hazards models, stratified by screening CD4 count and sex. Treatment discontinuation was ignored, including the initiation of statin therapy as part of clinical care (intention to treat policy).
Time Frame: as for outcome 1
Population: All participants enrolled according to the randomized treatment group.
Measure: Number (95% Confidence Interval); unit: events per 1000 person-years
Arm/Group | Pitavastatin | Placebo
Number analyzed (Participants) | 3888 | 3881
events per 1000 person-years | 9.31 [8.07 to 10.75] | 12.02 [10.60 to 13.63]
Statistical Analysis 1: Comparison: Pitavastatin vs Placebo; Test type: Superiority; Hazard Ratio (HR) = 0.77, 95% CI 2-sided [0.64 to 0.94] — Hazard ratio is shown as pitavastatin/placebo

11. Secondary Outcome: Incidence Rate of Death (All-cause)
Description: Death from any cause. The incidence rates were estimated based on time to event using Poisson distribution, with follow-up time censored at last contact. The treatment effect was estimated via relative hazard (i.e. hazard ratio) of prescribed pitavastatin compared to placebo from Cox proportional hazards models, stratified by screening CD4 count and sex. Treatment discontinuation was ignored, including the initiation of statin therapy as part of clinical care (intention to treat policy).
Time Frame: as for outcome 1
Population: All participants enrolled according to the randomized treatment group.
Measure: Number (95% Confidence Interval); unit: events per 1000 person-years
Arm/Group | Pitavastatin | Placebo
Number analyzed (Participants) | 3888 | 3881
events per 1000 person-years | 6.18 [5.19 to 7.36] | 6.99 [5.93 to 8.23]
Statistical Analysis 1: Comparison: Pitavastatin vs Placebo; Test type: Superiority; Hazard Ratio (HR) = 0.88, 95% CI 2-sided [0.70 to 1.12] — Hazard ratio is shown as pitavastatin/placebo

12. Secondary Outcome: Incidence Rate of Non-CV Clinical Diagnoses
Description: A composite of non-CV clinical diagnoses including: non-AIDS-defining cancers (excluding basal cell and squamous cell carcinomas of the skin), AIDS-defining events (based on Centers for Disease Control and Prevention [CDC] 2014 classification), end-stage renal disease, and end-stage liver disease. The incidence rates were estimated based on time to the first event using Poisson distribution, with follow-up time censored at last contact. The treatment effect was estimated via cause-specific relative hazard (i.e. hazard ratio) of prescribed pitavastatin compared to placebo from Cox proportional hazards models, stratified by screening CD4 count and sex. Deaths (without preceding event of interest) were treated as competing events and censored. Treatment discontinuation was ignored, including the initiation of statin therapy as part of clinical care (intention to treat policy).
Time Frame: as for outcome 1
Population: All participants enrolled according to the randomized treatment group.
Measure: Number (95% Confidence Interval); unit: events per 1000 person-years
Arm/Group | Pitavastatin | Placebo
Number analyzed (Participants) | 3888 | 3881
events per 1000 person-years | 9.17 [7.93 to 10.59] | 9.90 [8.61 to 11.38]
Statistical Analysis 1: Comparison: Pitavastatin vs Placebo; Test type: Superiority; Hazard Ratio (HR) = 0.92, 95% CI 2-sided [0.76 to 1.13] — Hazard ratio is shown as pitavastatin/placebo

13. Secondary Outcome: Incidence Rate of Non-AIDS-defining Cancer
Description: Non-AIDS-defining cancer (excluding basal cell and squamous cell carcinomas of the skin) component of the composite non-CV clinical diagnoses outcome. The incidence rates were estimated based on time to the first event using Poisson distribution, with follow-up time censored at last contact. The treatment effect was estimated via cause-specific relative hazard (i.e. hazard ratio) of prescribed pitavastatin compared to placebo from Cox proportional hazards models, stratified by screening CD4 count and sex. Deaths (without preceding event of interest) were treated as competing events and censored. Treatment discontinuation was ignored, including the initiation of statin therapy as part of clinical care (intention to treat policy).
Time Frame: as for outcome 1
Population: All participants enrolled according to the randomized treatment group.
Measure: Number (95% Confidence Interval); unit: events per 1000 person-years
Arm/Group | Pitavastatin | Placebo
Number analyzed (Participants) | 3888 | 3881
events per 1000 person-years | 5.25 [4.34 to 6.36] | 5.68 [4.74 to 6.83]
Statistical Analysis 1: Comparison: Pitavastatin vs Placebo; Test type: Superiority; Hazard Ratio (HR) = 0.93, 95% CI 2-sided [0.71 to 1.20] — Hazard ratio is shown as pitavastatin/placebo

14. Secondary Outcome: Incidence Rate of AIDS-defining Event
Description: AIDS-defining event component of the composite non-CV clinical diagnoses outcome. Events were captured based on the Centers for Disease Control and Prevention [CDC] 2014 classification. The incidence rates were estimated based on time to the first event using Poisson distribution, with follow-up time censored at last contact. The treatment effect was estimated via cause-specific relative hazard (i.e. hazard ratio) of prescribed pitavastatin compared to placebo from Cox proportional hazards models, stratified by screening CD4 count and sex. Deaths (without preceding event of interest) were treated as competing events and censored. Treatment discontinuation was ignored, including the initiation of statin therapy as part of clinical care (intention to treat policy).
Time Frame: as for outcome 1
Population: All participants enrolled according to the randomized treatment group.
Measure: Number (95% Confidence Interval); unit: events per 1000 person-years
Arm/Group | Pitavastatin | Placebo
Number analyzed (Participants) | 3888 | 3881
events per 1000 person-years | 3.36 [2.65 to 4.27] | 3.55 [2.82 to 4.47]
Statistical Analysis 1: Comparison: Pitavastatin vs Placebo; Test type: Superiority; Hazard Ratio (HR) = 0.94, 95% CI 2-sided [0.68 to 1.31] — Hazard ratio is shown as pitavastatin/placebo

15. Secondary Outcome: Incidence Rate of End-Stage Renal Disease
Description: End-stage renal disease (defined as initiation of dialysis or renal transplantation) component of the composite non-CV clinical diagnoses outcome. The incidence rates were estimated based on time to the first event using Poisson distribution, with follow-up time censored at last contact. The treatment effect was estimated via cause-specific relative hazard (i.e. hazard ratio) of prescribed pitavastatin compared to placebo from Cox proportional hazards models, stratified by screening CD4 count and sex. Deaths (without preceding event of interest) were treated as competing events and censored. Treatment discontinuation was ignored, including the initiation of statin therapy as part of clinical care (intention to treat policy).
Time Frame: as for outcome 1
Population: All participants enrolled according to the randomized treatment group.
Measure: Number (95% Confidence Interval); unit: events per 1000 person-years
Arm/Group | Pitavastatin | Placebo
Number analyzed (Participants) | 3888 | 3881
events per 1000 person-years | 0.15 [0.05 to 0.46] | 0.24 [0.10 to 0.59]
Statistical Analysis 1: Comparison: Pitavastatin vs Placebo; Test type: Superiority; Hazard Ratio (HR) = 0.60, 95% CI 2-sided [0.14 to 2.51] — Hazard ratio is shown as pitavastatin/placebo

16. Secondary Outcome: Incidence Rate of End-Stage Liver Disease
Description: End-stage liver disease (defined as cirrhosis or hepatic decompensation requiring hospitalization) component of the composite non-CV clinical diagnoses outcome. The incidence rates were estimated based on time to the first event using Poisson distribution, with follow-up time censored at last contact. The treatment effect was estimated via cause-specific relative hazard (i.e. hazard ratio) of prescribed pitavastatin compared to placebo from Cox proportional hazards models, stratified by screening CD4 count and sex. Deaths (without preceding event of interest) were treated as competing events and censored. Treatment discontinuation was ignored, including the initiation of statin therapy as part of clinical care (intention to treat policy).
Time Frame: as for outcome 1
Population: All participants enrolled according to the randomized treatment group.
Measure: Number (95% Confidence Interval); unit: events per 1000 person-years
Arm/Group | Pitavastatin | Placebo
Number analyzed (Participants) | 3888 | 3881
events per 1000 person-years | 0.59 [0.33 to 1.04] | 0.64 [0.37 to 1.10]
Statistical Analysis 1: Comparison: Pitavastatin vs Placebo; Test type: Superiority; Hazard Ratio (HR) = 0.92, 95% CI 2-sided [0.42 to 2.02] — Hazard ratio is shown as pitavastatin/placebo

17. Secondary Outcome: Incidence Rate of Non-fatal Serious Adverse Event
Description: Safety analysis outcome measure of non-fatal serious adverse event was defined by International Conference on Harmonisation (ICH) criteria. Fatal events were excluded as deaths were a secondary efficacy outcome (see outcome measure: incidence rate of death (all-cause)). The incidence rates were estimated based on time to the first event using Poisson distribution, with follow-up time censored at last contact. The treatment effect was estimated using incidence rate ratios from Poisson regression models (prescribed pitavastatin compared to placebo), adjusted for screening CD4 and sex. Treatment discontinuation was ignored, including the initiation of statin therapy as part of clinical care (intention to treat policy).
Time Frame: as for outcome 1
Population: All participants enrolled according to the randomized treatment group.
Measure: Number (95% Confidence Interval); unit: events per 100 person-years
Arm/Group | Pitavastatin | Placebo
Number analyzed (Participants) | 3888 | 3881
events per 100 person-years | 4.17 [3.88 to 4.48] | 4.18 [3.89 to 4.49]
Statistical Analysis 1: Comparison: Pitavastatin vs Placebo; Test type: Superiority; Incidence rate ratio = 1.00, 95% CI 2-sided [0.90 to 1.10] — Incidence rate ratio is shown as pitavastatin/placebo

18. Secondary Outcome: Incidence Rate of Diabetes
Description: Safety analysis outcome measure of diabetes was defined as new diagnosis of diabetes with initiation of anti-diabetic agent. The incidence rates were estimated based on time to the first event using Poisson distribution, with follow-up time censored at last contact. The treatment effect was estimated using incidence rate ratios from Poisson regression models (prescribed pitavastatin compared to placebo), adjusted for screening CD4 and sex. Treatment discontinuation was ignored, including the initiation of statin therapy as part of clinical care (intention to treat policy).
Time Frame: as for outcome 1
Population: Participants without pre-existing diabetes at baseline, according to the randomized treatment group.
Measure: Number (95% Confidence Interval); unit: events per 100 person-years
Arm/Group | Pitavastatin | Placebo
Number analyzed (Participants) | 3864 | 3867
events per 100 person-years | 1.18 [1.04 to 1.34] | 0.91 [0.79 to 1.06]
Statistical Analysis 1: Comparison: Pitavastatin vs Placebo; Test type: Superiority; Incidence rate ratio = 1.29, 95% CI 2-sided [1.07 to 1.57] — Incidence rate ratio is shown as pitavastatin/placebo

19. Secondary Outcome: Incidence Rate of Myalgia, Muscle Weakness or Myopathy
Description: Safety analysis outcome measure of myalgia, muscle weakness or myopathy which were grade 3 or higher or treatment-limiting. Grade 3 or higher includes grade 3 and 4 events, where grade 3 refers to severe and grade 4 to life-threatening according to DAIDS AE Grading Table (version 2.1). The incidence rates were estimated based on time to the first event using Poisson distribution, with follow-up time censored at last contact. The treatment effect was estimated using incidence rate ratios from Poisson regression models (prescribed pitavastatin compared to placebo), adjusted for screening CD4 and sex. Treatment discontinuation was ignored, including the initiation of statin therapy as part of clinical care (intention to treat policy).
Time Frame: as for outcome 1
Population: All participants enrolled according to the randomized treatment group.
Measure: Number (95% Confidence Interval); unit: events per 100 person-years
Arm/Group | Pitavastatin | Placebo
Number analyzed (Participants) | 3888 | 3881
events per 100 person-years | 0.46 [0.38 to 0.56] | 0.29 [0.23 to 0.38]
Statistical Analysis 1: Comparison: Pitavastatin vs Placebo; Test type: Superiority; Incidence rate ratio = 1.58, 95% CI 2-sided [1.14 to 2.19] — Incidence rate ratio is shown as pitavastatin/placebo

20. Secondary Outcome: Incidence Rate of Rhabdomyolysis
Description: Safety analysis outcome measure of rhabdomyolysis which was grade 3 or higher or treatment-limiting. Grade 3 or higher includes grade 3 and 4 events, where grade 3 refers to severe and grade 4 to life-threatening, according to DAIDS AE Grading Table (version 2.1). The incidence rates were estimated based on time to the first event using Poisson distribution, with follow-up time censored at last contact. The treatment effect was estimated using incidence rate ratios from Poisson regression models (prescribed pitavastatin compared to placebo). Due to small number of events, there was no adjustment for screening CD4 and sex. Treatment discontinuation was ignored, including the initiation of statin therapy as part of clinical care (intention to treat policy).
Time Frame: as for outcome 1
Population: All participants enrolled according to the randomized treatment group.
Measure: Number (95% Confidence Interval); unit: events per 100 person-years
Arm/Group | Pitavastatin | Placebo
Number analyzed (Participants) | 3888 | 3881
events per 100 person-years | 0.015 [0.005 to 0.046] | 0.020 [0.007 to 0.052]
Statistical Analysis 1: Comparison: Pitavastatin vs Placebo; Test type: Superiority; Incidence rate ratio = 0.75, 95% CI 2-sided [0.17 to 3.37] — Incidence rate ratio is shown as pitavastatin/placebo

21. Secondary Outcome: Incidence Rate of Grade 3 or Higher ALT
Description: Safety analysis outcome measure of Grade 3 or higher alanine transaminase (ALT). Grade 3 or higher includes grade 3 and 4 events, where grade 3 refers to severe and grade 4 to life-threatening, according to DAIDS AE Grading Table (version 2.1). The incidence rates were estimated based on time to the first event using Poisson distribution, with follow-up time censored at last contact. The treatment effect was estimated using incidence rate ratios from Poisson regression models (prescribed pitavastatin compared to placebo). Due to small number of events, there was no adjustment for screening CD4 and sex. Treatment discontinuation was ignored, including the initiation of statin therapy as part of clinical care (intention to treat policy).
Time Frame: as for outcome 1
Population: All participants enrolled according to the randomized treatment group.
Measure: Number (95% Confidence Interval); unit: events per 100 person-years
Arm/Group | Pitavastatin | Placebo
Number analyzed (Participants) | 3888 | 3881
events per 100 person-years | 0.059 [0.033 to 0.10] | 0.044 [0.023 to 0.085]
Statistical Analysis 1: Comparison: Pitavastatin vs Placebo; Test type: Superiority; Incidence rate ratio = 1.34, 95% CI 2-sided [0.56 to 3.18] — Incidence rate ratio is shown as pitavastatin/placebo

22. Secondary Outcome: Incidence Rate of Adverse Event (AE)
Description: Safety analysis outcome measure of any AE. AE collection included events of grade ≥3, those that were serious (defined by International Conference on Harmonisation (ICH) criteria) or treatment-limiting, and targeted diagnosis of diabetes. Grade ≥3 includes events that were grade 3 (serious) or grade 4 (life-threatening) per DAIDS AE Grading Table (version 2.1). Fatal events were excluded as deaths were a secondary efficacy outcome (see outcome measure: incidence rate of death (all-cause)). The incidence rates were estimated based on time to the first event using Poisson distribution, with follow-up time censored at last contact. The treatment effect was estimated using incidence rate ratios from Poisson regression models (prescribed pitavastatin compared to placebo), adjusted for screening CD4 and sex. Treatment discontinuation was ignored, including the initiation of statin therapy as part of clinical care (intention to treat policy).
Time Frame: as for outcome 1
Population: All participants enrolled according to the randomized treatment group.
Measure: Number (95% Confidence Interval); unit: events per 100 person-years
Arm/Group | Pitavastatin | Placebo
Number analyzed (Participants) | 3888 | 3881
events per 100 person-years | 8.83 [8.38 to 9.31] | 8.49 [8.05 to 8.95]
Statistical Analysis 1: Comparison: Pitavastatin vs Placebo; Test type: Superiority; Incidence rate ratio = 1.04, 95% CI 2-sided [0.97 to 1.12] — Incidence rate ratio is shown as pitavastatin/placebo

23. Secondary Outcome: Fasting Low-density Lipoprotein Cholesterol (LDL-C)
Description: LDL-C level was derived as LDL-C calculated according to the Friedewald formula at triglycerides ≤400 mg/dL, and direct LDL-C at triglycerides >400 to <500 mg/dL. Treatment discontinuation was ignored, including the initiation of statin therapy as part of clinical care (intention to treat policy).
Time Frame: At entry and months 12, 24, 36, 48, 60, 72, 84. Participants' follow-up time on study varied, depending on their time of enrollment.
Population: All participants enrolled according to the randomized treatment group. The number of participants with fasting LDL-C available is shown at each timepoint.
Measure: Median (Inter-Quartile Range); unit: mg/dL
Arm/Group | Pitavastatin | Placebo
Number analyzed (Participants) | 3888 | 3881
mg/dL
  Entry: LDL-C: number analyzed (Participants) | 3682 | 3667
  Entry: LDL-C | 107 [87 to 129] | 106 [86 to 127]
  Month 12: LDL-C: number analyzed (Participants) | 3341 | 3321
  Month 12: LDL-C | 74 [58 to 92] | 105 [85 to 126]
  Month 24: LDL-C: number analyzed (Participants) | 3088 | 3122
  Month 24: LDL-C | 75 [59 to 93] | 104 [84 to 126]
  Month 36: LDL-C: number analyzed (Participants) | 2810 | 2792
  Month 36: LDL-C | 73 [57 to 92] | 104 [83 to 126]
  Month 48: LDL-C: number analyzed (Participants) | 2525 | 2526
  Month 48: LDL-C | 73 [56 to 92] | 103 [83 to 124]
  Month 60: LDL-C: number analyzed (Participants) | 2057 | 2053
  Month 60: LDL-C | 73 [56 to 93] | 103 [82 to 125]
  Month 72: LDL-C: number analyzed (Participants) | 1170 | 1114
  Month 72: LDL-C | 74 [57 to 95] | 101 [82 to 122]
  Month 84: LDL-C: number analyzed (Participants) | 492 | 452
  Month 84: LDL-C | 75 [59 to 98] | 98 [81 to 121]

24. Secondary Outcome: Fasting Non-high-density Lipoprotein Cholesterol (Non-HDL-C)
Description: Non-HDL cholesterol levels were calculated as total cholesterol minus HDL cholesterol. Treatment discontinuation was ignored, including the initiation of statin therapy as part of clinical care (intention to treat policy).
Time Frame: as for outcome 23
Population: All participants enrolled according to the randomized treatment group. The number of participants with fasting non-HDL-C available is shown at each timepoint.
Measure: Median (Inter-Quartile Range); unit: mg/dL
Arm/Group | Pitavastatin | Placebo
Number analyzed (Participants) | 3888 | 3881
mg/dL
  Entry: non-HDL-C: number analyzed (Participants) | 3714 | 3681
  Entry: non-HDL-C | 133 [110 to 158] | 132 [108 to 157]
  Month 12: non-HDL-C: number analyzed (Participants) | 3367 | 3354
  Month 12: non-HDL-C | 97 [80 to 118] | 131 [108 to 156]
  Month 24: non-HDL-C: number analyzed (Participants) | 3116 | 3143
  Month 24: non-HDL-C | 98 [80 to 121] | 131 [108 to 156]
  Month 36: non-HDL-C: number analyzed (Participants) | 2835 | 2816
  Month 36: non-HDL-C | 97 [78 to 118] | 130 [107 to 154]
  Month 48: non-HDL-C: number analyzed (Participants) | 2542 | 2544
  Month 48: non-HDL-C | 96 [77 to 119] | 128 [106 to 154]
  Month 60: non-HDL-C: number analyzed (Participants) | 2073 | 2074
  Month 60: non-HDL-C | 96 [78 to 120] | 127 [104 to 153]
  Month 72: non-HDL-C: number analyzed (Participants) | 1180 | 1121
  Month 72: non-HDL-C | 95 [78 to 121] | 124 [104 to 150]
  Month 84: non-HDL-C: number analyzed (Participants) | 496 | 455
  Month 84: non-HDL-C | 99 [80 to 124] | 123 [101 to 151]

25. Secondary Outcome: Incidence Rate of Serious COVID-19
Description: Serious COVID-19 was defined as COVID-19 that resulted in hospitalization or death or was life-threatening as per the International Conference on Harmonisation of Technical Requirements for Registration of Pharmaceuticals for Human Use Guideline E2A definition. The incidence rates were estimated based on time to the first event using Poisson distribution, with follow-up time censored at last contact. The treatment effect was estimated using incidence rate ratios from Poisson regression models (prescribed pitavastatin compared to placebo), adjusted for GBD region to account for regional differences. Treatment discontinuation was ignored, including the initiation of statin therapy as part of clinical care (intention to treat policy).
Time Frame: From January 1, 2020 through end of study; the median follow-up time was 3.3 years.
Population: Participants who remained in REPRIEVE follow-up at the start of the COVID-19 pandemic (defined as January 1, 2020), according to the randomized treatment group.
Measure: Number (95% Confidence Interval); unit: events per 100 person-years
Arm/Group | Pitavastatin | Placebo
Number analyzed (Participants) | 3451 | 3454
events per 100 person-years | 0.45 [0.34 to 0.59] | 0.60 [0.48 to 0.77]
Statistical Analysis 1: Comparison: Pitavastatin vs Placebo; Test type: Superiority; Incidence rate ratio = 0.75, 95% CI 2-sided [0.52 to 1.08] — Incidence rate ratio is shown as pitavastatin/placebo

26. Secondary Outcome: Incidence Rate of COVID-19
Description: COVID-19 was defined as COVID-19 clinical diagnosis or positive test result (SARS-CoV-2 PCR or rapid antigen tests). The incidence rates were estimated based on time to the first event using Poisson distribution, with follow-up time censored at last contact. The treatment effect was estimated using incidence rate ratios (prescribed pitavastatin compared to placebo) from Poisson regression models, adjusted for GBD region to account for regional differences. Treatment discontinuation was ignored, including the initiation of statin therapy as part of clinical care (intention to treat policy).
Time Frame: From January 1, 2020 through end of study; the median follow-up time was 3.3 years.
Population: as for outcome 25
Measure: Number (95% Confidence Interval); unit: events per 100 person-years
Arm/Group | Pitavastatin | Placebo
Number analyzed (Participants) | 3451 | 3454
events per 100 person-years | 8.79 [8.22 to 9.39] | 8.35 [7.80 to 8.93]
Statistical Analysis 1: Comparison: Pitavastatin vs Placebo; Test type: Superiority; Incidence rate ratio = 1.05, 95% CI 2-sided [0.96 to 1.16] — Incidence rate ratio is shown as pitavastatin/placebo

27. Secondary Outcome: For Mechanistic Substudy: Change in Non-Calcified Plaque (NCP) Volume From Baseline to Year 2
Description: NCP was defined as plaque voxels with attenuation of <350. Change in NCP is expressed as absolute change from baseline (calculated as NCP volume at 2 years minus NCP volume at entry), based on quantitative read of the CT scan, whenever available. Participants without a quantitative read and no evidence of NCP based on the corresponding qualitative read were assigned a value of zero for the change. Treatment discontinuation was ignored, including the initiation of statin therapy as part of clinical care (intention to treat policy).
Time Frame: Entry and Year 2.
Population: Participants enrolled in the Mechanistic Substudy, with complete case outcome data (paired entry and year 2).
Measure: Mean (Standard Deviation); unit: mm^3
Groups:
- Pitavastatin (Substudy): Participants enrolled in the Mechanistic Substudy randomized to pitavastatin in the parent study. In the parent study, participants received pitavastatin once a day for the entire time they were in study follow-up.
  Pitavastatin: One tablet (4 mg) taken once daily, orally with or without food
- Placebo (Substudy): Participants enrolled in the Mechanistic Substudy randomized to placebo in the parent study. In the parent study, participants received placebo for pitavastatin once a day for the entire time they were in study follow-up.
  Placebo: One tablet taken once daily, orally with or without food
Arm/Group | Pitavastatin (Substudy) | Placebo (Substudy)
Number analyzed (Participants) | 290 | 297
mm^3 | -1.70 (25.2) | 2.62 (27.1)
Statistical Analysis 1: Comparison: Pitavastatin (Substudy) vs Placebo (Substudy); Test type: Superiority; p = 0.04, Regression, Linear; Mean Difference (Net) = -4.3, 95% CI 2-sided [-8.6 to -0.1] — Treatment group difference was estimated as baseline-adjusted mean difference in change at year 2, using linear regression

28. Secondary Outcome: For Mechanistic Substudy: Number of Participants With Progression of NCP From Baseline to Year 2
Description: Progression at Year 2 was defined as any progression/increase in NCP volume in participants with evidence of NCP at entry, or incident NCP in participants without evidence of NCP at entry. Treatment discontinuation was ignored, including the initiation of statin therapy as part of clinical care (intention to treat policy).
Time Frame: Entry and year 2.
Population: Participants enrolled in the Mechanistic Substudy, with complete case outcome data (paired entry and year 2).
Measure: Count of Participants; unit: Participants
Arm/Group | Pitavastatin (Substudy) | Placebo (Substudy)
Number analyzed (Participants) | 302 | 309
Participants | 53 | 85
Statistical Analysis 1: Comparison: Pitavastatin (Substudy) vs Placebo (Substudy); Test type: Superiority; p = 0.003, Chi-squared; Risk Ratio (RR) = 0.67, 95% CI 2-sided [0.52 to 0.88] — Treatment effect was estimated as relative risk (pitavastatin/placebo), adjusted for presence of NCP at entry

29. Secondary Outcome: For Mechanistic Substudy: Change in Total Plaque Volume From Baseline to Year 2
Description: Total plaque includes all plaque voxels (noncalcified + calcified). Change in total plaque volume is expressed as absolute change from baseline (calculated as volume at 2 years minus volume at entry). Treatment discontinuation was ignored, including the initiation of statin therapy as part of clinical care (intention to treat policy).
Time Frame: Entry and year 2.
Population: Participants enrolled in the Mechanistic Substudy, with complete case outcome data (paired entry and year 2).
Measure: Mean (Standard Deviation); unit: mm^3
Arm/Group | Pitavastatin (Substudy) | Placebo (Substudy)
Number analyzed (Participants) | 302 | 309
mm^3 | 2.34 (28.7) | 6.89 (32.3)
Statistical Analysis 1: Comparison: Pitavastatin (Substudy) vs Placebo (Substudy); Test type: Superiority; Mean Difference (Net) = -4.3, 95% CI 2-sided [-9.2 to 0.62] — Treatment group difference was estimated as baseline-adjusted difference in mean change at year 2, using linear regression

30. Secondary Outcome: For Mechanistic Substudy: LpPLA2 Level
Description: Level of inflammatory biomarker lipoprotein-associated phospholipase A2 (LpPLA2). Treatment discontinuation was ignored, including the initiation of statin therapy as part of clinical care (intention to treat policy).
Time Frame: Entry and month 24.
Population: Participants enrolled in the Mechanistic Substudy with biomarker results available.
Measure: Median (Inter-Quartile Range); unit: ng/mL
Arm/Group | Pitavastatin (Substudy) | Placebo (Substudy)
Number analyzed (Participants) | 402 | 402
ng/mL
  Entry: number analyzed (Participants) | 398 | 391
  Entry | 126 [94.8 to 169] | 131 [89.6 to 163]
  Month 24: number analyzed (Participants) | 335 | 333
  Month 24 | 119 [84.0 to 160] | 143 [105 to 186]
Statistical Analysis 1: Comparison: Pitavastatin (Substudy) vs Placebo (Substudy); Comparison of LpPla2 Levels at Month 24; Test type: Superiority; p < 0.001, Wilcoxon (Mann-Whitney)

31. Secondary Outcome: For Mechanistic Substudy: Change in LpPLA2 From Baseline
Description: Change in inflammatory biomarker LpPLA2 from baseline calculated as value at month 24 minus value at entry. Treatment discontinuation was ignored, including the initiation of statin therapy as part of clinical care (intention to treat policy).
Time Frame: Entry and month 24.
Population: Participants enrolled in the Mechanistic Substudy with biomarker results available at entry and month 24.
Measure: Median (Inter-Quartile Range); unit: ng/mL
Arm/Group | Pitavastatin (Substudy) | Placebo (Substudy)
Number analyzed (Participants) | 335 | 333
ng/mL | -9.77 [-33.6 to 16.8] | 19.9 [-5.6 to 43.0]
Statistical Analysis 1: Comparison: Pitavastatin (Substudy) vs Placebo (Substudy); Comparison of Change in LpPla2 from Baseline at Month 24; Test type: Superiority; p < 0.001, Wilcoxon (Mann-Whitney)

32. Secondary Outcome: For Mechanistic Substudy: HsCRP Level
Description: Level of inflammatory marker high-sensitivity C-reactive protein (HsCRP). Censored values below or above the assay limit were imputed. Treatment discontinuation was ignored, including the initiation of statin therapy as part of clinical care (intention to treat policy).
Time Frame: Entry and month 24.
Population: Participants enrolled in the Mechanistic Substudy with biomarker results available.
Measure: Median (Inter-Quartile Range); unit: mg/dL
Arm/Group | Pitavastatin (Substudy) | Placebo (Substudy)
Number analyzed (Participants) | 402 | 402
mg/dL
  Entry: number analyzed (Participants) | 397 | 391
  Entry | 0.18 [0.08 to 0.39] | 0.18 [0.09 to 0.33]
  Month 24: number analyzed (Participants) | 343 | 335
  Month 24 | 0.17 [0.07 to 0.36] | 0.19 [0.10 to 0.40]
Statistical Analysis 1: Comparison: Pitavastatin (Substudy) vs Placebo (Substudy); Comparison of hsCRP Levels at Month 24; Test type: Superiority; p = 0.02, Wilcoxon (Mann-Whitney)

33. Secondary Outcome: For Mechanistic Substudy: Change in HsCRP From Baseline
Description: Change in inflammatory biomarker hsCRP from baseline calculated as value at month 24 minus value at entry. Treatment discontinuation was ignored, including the initiation of statin therapy as part of clinical care (intention to treat policy).
Time Frame: Entry and month 24.
Population: Participants enrolled in the Mechanistic Substudy with biomarker results available at entry and month 24.
Measure: Median (Inter-Quartile Range); unit: mg/mL
Arm/Group | Pitavastatin (Substudy) | Placebo (Substudy)
Number analyzed (Participants) | 343 | 335
mg/mL | -0.01 [-0.10 to 0.08] | 0.01 [-0.09 to 0.11]
Statistical Analysis 1: Comparison: Pitavastatin (Substudy) vs Placebo (Substudy); Comparison of Change in hsCRP from Baseline at Month 24; Test type: Superiority; p = 0.09, Wilcoxon (Mann-Whitney)

34. Secondary Outcome: For Mechanistic Substudy: Soluble CD163 Level
Description: Level of immune biomarker soluble CD163. Treatment discontinuation was ignored, including the initiation of statin therapy as part of clinical care (intention to treat policy).
Time Frame: Entry and month 24.
Population: Participants enrolled in the Mechanistic Substudy with biomarker results available.
Measure: Median (Inter-Quartile Range); unit: ng/mL
Arm/Group | Pitavastatin (Substudy) | Placebo (Substudy)
Number analyzed (Participants) | 402 | 402
ng/mL
  Entry: number analyzed (Participants) | 398 | 391
  Entry | 849 [651 to 1163] | 845 [613 to 1074]
  Month 24: number analyzed (Participants) | 335 | 333
  Month 24 | 1013 [728 to 1419] | 1003 [745 to 1384]
Statistical Analysis 1: Comparison: Pitavastatin (Substudy) vs Placebo (Substudy); Comparison of soluble CD163 Levels at Month 24; Test type: Superiority; p = 0.65, Wilcoxon (Mann-Whitney)

35. Secondary Outcome: For Mechanistic Substudy: Change in Soluble CD163 From Baseline
Description: Change in immune biomarker soluble CD163 from baseline calculated as value at month 24 minus value at entry. Treatment discontinuation was ignored, including the initiation of statin therapy as part of clinical care (intention to treat policy).
Time Frame: Entry and month 24.
Population: Participants enrolled in the Mechanistic Substudy with biomarker results available at entry and month 24.
Measure: Median (Inter-Quartile Range); unit: ng/mL
Arm/Group | Pitavastatin (Substudy) | Placebo (Substudy)
Number analyzed (Participants) | 335 | 330
ng/mL | 149 [-60.8 to 420] | 143 [-46.0 to 453]
Statistical Analysis 1: Comparison: Pitavastatin (Substudy) vs Placebo (Substudy); Comparison of Change in soluble CD163 from Baseline at Month 24; Test type: Superiority; p = 0.88, Wilcoxon (Mann-Whitney)

36. Other Pre Specified Outcome: Incidence Rate of MACE by Sex
Description: Subgroup analysis of the primary composite MACE outcome measure (as described above) by sex. The incidence rates were estimated based on time to the first event using Poisson distribution, with follow-up time censored at last contact. The Cox proportional hazards models described for the primary outcome above were expanded to include sex and interaction of sex and treatment, to evaluate modification of statin effect.
Time Frame: as for outcome 1
Population: All participants enrolled according to the randomized treatment group.
Measure: Number (95% Confidence Interval); unit: events per 1000 person-years
Arm/Group | Pitavastatin | Placebo
Number analyzed (Participants) | 3888 | 3881
events per 1000 person-years
  Among females: number analyzed (Participants) | 1211 | 1208
  Among females | 3.9 [2.7 to 5.8] | 6.2 [4.6 to 8.4]
  Among males: number analyzed (Participants) | 2677 | 2673
  Among males | 5.5 [4.4 to 6.9] | 8.5 [7.1 to 10.2]
Statistical Analysis 1: Comparison: Pitavastatin vs Placebo; Evaluation of treatment effect modification by sex (i.e. pitavastatin effect differing in females compared to males); Test type: Superiority; p = 0.98, Regression, Cox; Treatment effect modification by sex was evaluated via interaction of treatment and sex in the Cox proportional hazards regression model
Statistical Analysis 2: Comparison: Pitavastatin vs Placebo; Evaluation of pitavastatin effect among females; Test type: Superiority; Hazard Ratio (HR) = 0.63, 95% CI 2-sided [0.39 to 1.04] — Hazard ratio is shown as pitavastatin/placebo among females
Statistical Analysis 3: Comparison: Pitavastatin vs Placebo; Evaluation of pitavastatin effect among males; Test type: Superiority; Hazard Ratio (HR) = 0.64, 95% CI 2-sided [0.48 to 0.86] — Hazard ratio is shown as pitavastatin/placebo among males

37. Other Pre Specified Outcome: Incidence Rate of MACE by Race
Description: Subgroup analysis of the primary composite MACE outcome measure (as described above) by race. The incidence rates were estimated based on time to the first event using Poisson distribution, with follow-up time censored at last contact. The Cox proportional hazards models described for the primary outcome above were expanded to include race and interaction of race and treatment, to evaluate modification of statin effect.
Time Frame: as for outcome 1
Population: All participants enrolled according to the randomized treatment group.
Measure: Number (95% Confidence Interval); unit: events per 1000 person-years
Arm/Group | Pitavastatin | Placebo
Number analyzed (Participants) | 3888 | 3881
events per 1000 person-years
  Among Asians: number analyzed (Participants) | 571 | 567
  Among Asians | 1.6 [0.7 to 3.7] | 7.0 [4.6 to 10.6]
  Among Blacks: number analyzed (Participants) | 1569 | 1639
  Among Blacks | 5.8 [4.3 to 7.7] | 8.7 [6.9 to 10.9]
  Among Whites: number analyzed (Participants) | 1364 | 1340
  Among Whites | 5.6 [4.1 to 7.7] | 7.5 [5.7 to 9.9]
  Among Other: number analyzed (Participants) | 384 | 335
  Among Other | 5.0 [2.7 to 9.4] | 5.7 [3.1 to 10.6]
Statistical Analysis 1: Comparison: Pitavastatin vs Placebo; Evaluation of treatment effect modification by race (i.e. pitavastatin effect differing between races); Test type: Superiority; p = 0.14, Regression, Cox; Treatment effect modification by race was evaluated via interaction of treatment and race in the Cox proportional hazards regression model
Statistical Analysis 2: Comparison: Pitavastatin vs Placebo; Pitavastatin effect among Asians from subgroup analysis by race; Test type: Superiority; Hazard Ratio (HR) = 0.22, 95% CI 2-sided [0.09 to 0.59]; Hazard ratio is shown as pitavastatin/placebo among Asians
Statistical Analysis 3: Comparison: Pitavastatin vs Placebo; Pitavastatin effect among Blacks from subgroup analysis by race; Test type: Superiority; Hazard Ratio (HR) = 0.66, 95% CI 2-sided [0.46 to 0.96] — Hazard ratio is shown as pitavastatin/placebo among Blacks
Statistical Analysis 4: Comparison: Pitavastatin vs Placebo; Pitavastatin effect among Whites from subgroup analysis by race; Test type: Superiority; Hazard Ratio (HR) = 0.74, 95% CI 2-sided [0.49 to 1.13] — Hazard ratio is shown as pitavastatin/placebo among Whites
Statistical Analysis 5: Comparison: Pitavastatin vs Placebo; Pitavastatin effect among Other race from subgroup analysis by race; Test type: Superiority; Hazard Ratio (HR) = 0.87, 95% CI 2-sided [0.36 to 2.10]; Hazard ratio is shown as pitavastatin/placebo among Other race

ADVERSE EVENTS:
Time Frame: From entry through end of study. Follow-up time varied depending on time of enrollment (the median follow-up time was 5.6 years).
Description: AE collection included events of grade ≥3, those that were serious (per ICH criteria) or treatment-limiting, and all new diagnoses of diabetes. Grade ≥3 includes events that were grade 3 (serious) or grade 4 (life-threatening) per DAIDS AE Grading Table (version 2.1). Targeted clinical events for pitavastatin efficacy evaluation (MACE, death, COVID-19, heart failure) were not considered AEs. MedDRA High Level Term (HLT) grouped by System Organ Class is presented in the summary tables.
Arm/Group | Pitavastatin | Placebo
All-Cause Mortality (participants affected / at risk) | 126/3888 | 143/3881
Serious Adverse Events (participants affected / at risk) | 750/3888 | 755/3881
Other Adverse Events (participants affected / at risk) | 488/3888 | 420/3881
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pitavastatin (N=3888) | Placebo (N=3881)
Anaemia deficiencies (Blood and lymphatic system disorders) | 2 | 3
Anaemias NEC (Blood and lymphatic system disorders) | 16 | 10
Anaemias due to chronic disorders (Blood and lymphatic system disorders) | 1 | 0
Coagulopathies (Blood and lymphatic system disorders) | 0 | 1
Leukopenias NEC (Blood and lymphatic system disorders) | 1 | 2
Lymphatic system disorders NEC (Blood and lymphatic system disorders) | 2 | 1
Neutropenias (Blood and lymphatic system disorders) | 2 | 2
Thrombocytopenias (Blood and lymphatic system disorders) | 3 | 4
Cardiac conduction disorders (Cardiac disorders) | 1 | 0
Cardiac signs and symptoms NEC (Cardiac disorders) | 0 | 1
Coronary artery disorders NEC (Cardiac disorders) | 1 | 0
Heart failures NEC (Cardiac disorders) | 5 | 6
Ischaemic coronary artery disorders (Cardiac disorders) | 7 | 10
Left ventricular failures (Cardiac disorders) | 2 | 1
Mitral valvular disorders (Cardiac disorders) | 1 | 0
Noninfectious pericarditis (Cardiac disorders) | 1 | 1
Pericardial disorders NEC (Cardiac disorders) | 1 | 3
Rate and rhythm disorders NEC (Cardiac disorders) | 3 | 2
Supraventricular arrhythmias (Cardiac disorders) | 8 | 6
Ventricular arrhythmias and cardiac arrest (Cardiac disorders) | 1 | 3
Hearing losses (Ear and labyrinth disorders) | 1 | 0
Inner ear signs and symptoms (Ear and labyrinth disorders) | 1 | 7
Adrenal cortical hypofunctions (Endocrine disorders) | 4 | 0
Hyperparathyroid disorders (Endocrine disorders) | 1 | 0
Posterior pituitary disorders (Endocrine disorders) | 0 | 2
Cataract conditions (Eye disorders) | 12 | 6
Choroid and vitreous structural change, deposit and degeneration (Eye disorders) | 2 | 0
Glaucomas (excl congenital) (Eye disorders) | 1 | 0
Iris and uveal tract infections, irritations and inflammations (Eye disorders) | 1 | 0
Optic disc abnormalities NEC (Eye disorders) | 1 | 0
Optic nerve bleeding and vascular disorders (Eye disorders) | 1 | 0
Orbital infections, inflammations and irritations (Eye disorders) | 0 | 1
Retinal structural change, deposit and degeneration (Eye disorders) | 3 | 1
Visual impairment and blindness (excl colour blindness) (Eye disorders) | 3 | 0
Abdominal hernias NEC (Gastrointestinal disorders) | 3 | 2
Acute and chronic pancreatitis (Gastrointestinal disorders) | 10 | 11
Anal and rectal disorders NEC (Gastrointestinal disorders) | 1 | 1
Anal and rectal pains (Gastrointestinal disorders) | 2 | 0
Benign neoplasms gastrointestinal (excl oral cavity) (Gastrointestinal disorders) | 0 | 1
Colitis (excl infective) (Gastrointestinal disorders) | 4 | 8
Diaphragmatic hernias (Gastrointestinal disorders) | 0 | 2
Diarrhoea (excl infective) (Gastrointestinal disorders) | 9 | 4
Duodenal and small intestinal stenosis and obstruction (Gastrointestinal disorders) | 4 | 2
Duodenal ulcers and perforation (Gastrointestinal disorders) | 1 | 0
Gastric and oesophageal haemorrhages (Gastrointestinal disorders) | 0 | 2
Gastritis (excl infective) (Gastrointestinal disorders) | 8 | 2
Gastrointestinal and abdominal pains (excl oral and throat) (Gastrointestinal disorders) | 5 | 2
Gastrointestinal atonic and hypomotility disorders NEC (Gastrointestinal disorders) | 3 | 4
Gastrointestinal disorders NEC (Gastrointestinal disorders) | 0 | 1
Gastrointestinal inflammatory disorders NEC (Gastrointestinal disorders) | 1 | 3
Gastrointestinal signs and symptoms NEC (Gastrointestinal disorders) | 4 | 1
Gastrointestinal stenosis and obstruction NEC (Gastrointestinal disorders) | 5 | 4
Gastrointestinal ulcers and perforation, site unspecified (Gastrointestinal disorders) | 1 | 0
Gastrointestinal vascular occlusion and infarction (Gastrointestinal disorders) | 0 | 1
Gingival disorders, signs and symptoms NEC (Gastrointestinal disorders) | 0 | 1
Haemorrhoids and gastrointestinal varices (excl oesophageal) (Gastrointestinal disorders) | 2 | 1
Inguinal hernias (Gastrointestinal disorders) | 8 | 4
Intestinal haemorrhages (Gastrointestinal disorders) | 2 | 0
Intestinal ulcers and perforation NEC (Gastrointestinal disorders) | 1 | 4
Large intestinal stenosis and obstruction (Gastrointestinal disorders) | 1 | 0
Nausea and vomiting symptoms (Gastrointestinal disorders) | 8 | 1
Non-site specific gastrointestinal haemorrhages (Gastrointestinal disorders) | 2 | 11
Oesophageal stenosis and obstruction (Gastrointestinal disorders) | 1 | 0
Oesophageal ulcers and perforation (Gastrointestinal disorders) | 1 | 1
Oesophagitis (excl infective) (Gastrointestinal disorders) | 0 | 2
Oral soft tissue disorders NEC (Gastrointestinal disorders) | 0 | 1
Peritoneal and retroperitoneal disorders (Gastrointestinal disorders) | 2 | 0
Rectal inflammations NEC (Gastrointestinal disorders) | 2 | 0
Salivary gland disorders NEC (Gastrointestinal disorders) | 1 | 0
Umbilical hernias (Gastrointestinal disorders) | 3 | 1
Asthenic conditions (General disorders) | 1 | 0
Body temperature altered (General disorders) | 1 | 1
Febrile disorders (General disorders) | 5 | 4
General signs and symptoms NEC (General disorders) | 1 | 0
Healing abnormal NEC (General disorders) | 1 | 0
Hernias NEC (General disorders) | 0 | 1
Inflammations (General disorders) | 2 | 1
Oedema NEC (General disorders) | 1 | 0
Pain and discomfort NEC (General disorders) | 16 | 24
Ulcers NEC (General disorders) | 1 | 0
Bile duct infections and inflammations (Hepatobiliary disorders) | 0 | 3
Cholecystitis and cholelithiasis (Hepatobiliary disorders) | 17 | 13
Cholestasis and jaundice (Hepatobiliary disorders) | 0 | 1
Hepatic and hepatobiliary disorders NEC (Hepatobiliary disorders) | 1 | 1
Hepatic enzymes and function abnormalities (Hepatobiliary disorders) | 1 | 0
Hepatic fibrosis and cirrhosis (Hepatobiliary disorders) | 1 | 1
Hepatic vascular disorders (Hepatobiliary disorders) | 2 | 1
Hepatocellular damage and hepatitis NEC (Hepatobiliary disorders) | 0 | 4
Obstructive bile duct disorders (excl neoplasms) (Hepatobiliary disorders) | 1 | 3
Structural and other bile duct disorders (Hepatobiliary disorders) | 0 | 1
Acute and chronic sarcoidosis (Immune system disorders) | 0 | 1
Allergic conditions NEC (Immune system disorders) | 0 | 2
Allergies to foods, food additives, drugs and other chemicals (Immune system disorders) | 1 | 0
Anaphylactic and anaphylactoid responses (Immune system disorders) | 1 | 1
Abdominal and gastrointestinal infections (Infections and infestations) | 36 | 41
Actinomycotic infectious disorders (Infections and infestations) | 1 | 0
Adenoviral infections (Infections and infestations) | 0 | 1
Atypical mycobacterial infections (Infections and infestations) | 1 | 1
Bacterial infections NEC (Infections and infestations) | 41 | 30
Bone and joint infections (Infections and infestations) | 9 | 9
Breast infections (Infections and infestations) | 2 | 0
Caliciviral infections (Infections and infestations) | 0 | 1
Campylobacter infections (Infections and infestations) | 1 | 0
Candida infections (Infections and infestations) | 1 | 1
Central nervous system and spinal infections (Infections and infestations) | 5 | 2
Clostridia infections (Infections and infestations) | 5 | 2
Cryptococcal infections (Infections and infestations) | 1 | 0
Cytomegaloviral infections (Infections and infestations) | 0 | 1
Dental and oral soft tissue infections (Infections and infestations) | 3 | 1
Ear infections (Infections and infestations) | 0 | 2
Enterococcal infections (Infections and infestations) | 0 | 1
Escherichia infections (Infections and infestations) | 4 | 6
Eye and eyelid infections (Infections and infestations) | 2 | 0
Female reproductive tract infections (Infections and infestations) | 2 | 2
Flaviviral infections (Infections and infestations) | 6 | 9
Fungal infections NEC (Infections and infestations) | 1 | 0
Haemophilus infections (Infections and infestations) | 1 | 0
Hepatitis virus infections (Infections and infestations) | 3 | 6
Hepatobiliary and spleen infections (Infections and infestations) | 1 | 2
Herpes viral infections (Infections and infestations) | 7 | 7
Infections NEC (Infections and infestations) | 11 | 16
Influenza viral infections (Infections and infestations) | 11 | 10
Legionella infections (Infections and infestations) | 0 | 3
Leptospira infections (Infections and infestations) | 0 | 1
Listeria infections (Infections and infestations) | 0 | 1
Lower respiratory tract and lung infections (Infections and infestations) | 71 | 66
Male reproductive tract infections (Infections and infestations) | 4 | 7
Muscle and soft tissue infections (Infections and infestations) | 2 | 3
Neisseria infections (Infections and infestations) | 1 | 1
Nematode infections (Infections and infestations) | 1 | 0
Orthopox viral infections (Infections and infestations) | 1 | 2
Parainfluenzae viral infections (Infections and infestations) | 2 | 1
Plasmodia infections (Infections and infestations) | 1 | 0
Pneumocystis infections (Infections and infestations) | 2 | 2
Rhinoviral infections (Infections and infestations) | 2 | 0
Rickettsial infectious disorders NEC (Infections and infestations) | 2 | 0
Salmonella infections (Infections and infestations) | 2 | 0
Sepsis, bacteraemia, viraemia and fungaemia NEC (Infections and infestations) | 20 | 18
Shigella infections (Infections and infestations) | 0 | 1
Skin structures and soft tissue infections (Infections and infestations) | 1 | 3
Staphylococcal infections (Infections and infestations) | 4 | 4
Streptococcal infections (Infections and infestations) | 6 | 1
Toxoplasma infections (Infections and infestations) | 1 | 1
Treponema infections (Infections and infestations) | 6 | 10
Tuberculous infections (Infections and infestations) | 11 | 13
Upper respiratory tract infections (Infections and infestations) | 4 | 5
Urinary tract infections (Infections and infestations) | 23 | 15
Vascular infections (Infections and infestations) | 1 | 0
Viral infections NEC (Infections and infestations) | 5 | 8
Abdominal and gastrointestinal injuries NEC (Injury, poisoning and procedural complications) | 2 | 3
Accidental exposures to product (Injury, poisoning and procedural complications) | 0 | 1
Cerebral injuries NEC (Injury, poisoning and procedural complications) | 10 | 8
Chemical injuries (Injury, poisoning and procedural complications) | 0 | 1
Chest and respiratory tract injuries NEC (Injury, poisoning and procedural complications) | 4 | 1
Conditions caused by cold (Injury, poisoning and procedural complications) | 0 | 1
Eye injuries NEC (Injury, poisoning and procedural complications) | 1 | 2
Fractures and dislocations NEC (Injury, poisoning and procedural complications) | 7 | 3
Gastrointestinal and hepatobiliary procedural complications (Injury, poisoning and procedural complications) | 2 | 0
Limb fractures and dislocations (Injury, poisoning and procedural complications) | 43 | 50
Muscle, tendon and ligament injuries (Injury, poisoning and procedural complications) | 3 | 0
Musculoskeletal procedural complications (Injury, poisoning and procedural complications) | 0 | 1
Non-site specific injuries NEC (Injury, poisoning and procedural complications) | 14 | 12
Non-site specific procedural complications (Injury, poisoning and procedural complications) | 2 | 7
Overdoses NEC (Injury, poisoning and procedural complications) | 4 | 4
Pelvic fractures and dislocations (Injury, poisoning and procedural complications) | 1 | 1
Poisoning and toxicity (Injury, poisoning and procedural complications) | 3 | 3
Product administration errors and issues (Injury, poisoning and procedural complications) | 0 | 4
Radiation injuries (Injury, poisoning and procedural complications) | 0 | 1
Site specific injuries NEC (Injury, poisoning and procedural complications) | 3 | 5
Skin injuries NEC (Injury, poisoning and procedural complications) | 1 | 2
Skull fractures, facial bone fractures and dislocations (Injury, poisoning and procedural complications) | 1 | 3
Spinal cord injuries NEC (Injury, poisoning and procedural complications) | 1 | 0
Spinal fractures and dislocations (Injury, poisoning and procedural complications) | 4 | 3
Thermal burns (Injury, poisoning and procedural complications) | 3 | 2
Thoracic cage fractures and dislocations (Injury, poisoning and procedural complications) | 6 | 3
Carbohydrate tolerance analyses (incl diabetes) (Investigations) | 2 | 0
Cardiac function diagnostic procedures (Investigations) | 0 | 1
ECG investigations (Investigations) | 0 | 1
Hepatobiliary function diagnostic procedures (Investigations) | 8 | 4
Physical examination procedures and organ system status (Investigations) | 0 | 4
Platelet analyses (Investigations) | 1 | 0
Red blood cell analyses (Investigations) | 2 | 1
Renal function analyses (Investigations) | 4 | 5
Skeletal and cardiac muscle analyses (Investigations) | 1 | 1
Tissue enzyme analyses NEC (Investigations) | 0 | 1
Triglyceride analyses (Investigations) | 2 | 1
Vascular tests NEC (incl blood pressure) (Investigations) | 3 | 3
White blood cell analyses (Investigations) | 1 | 2
Calcium metabolism disorders (Metabolism and nutrition disorders) | 1 | 1
Diabetes mellitus (incl subtypes) (Metabolism and nutrition disorders) | 3 | 11
Diabetic complications NEC (Metabolism and nutrition disorders) | 2 | 4
Diabetic complications neurological (Metabolism and nutrition disorders) | 1 | 0
Disorders of purine metabolism (Metabolism and nutrition disorders) | 3 | 1
Elevated triglycerides (Metabolism and nutrition disorders) | 1 | 0
General nutritional disorders NEC (Metabolism and nutrition disorders) | 7 | 6
Hyperglycaemic conditions NEC (Metabolism and nutrition disorders) | 4 | 3
Hypoglycaemic conditions NEC (Metabolism and nutrition disorders) | 2 | 1
Lipid metabolism and deposit disorders NEC (Metabolism and nutrition disorders) | 0 | 1
Metabolic acidoses (excl diabetic acidoses) (Metabolism and nutrition disorders) | 2 | 3
Metabolic alkaloses (Metabolism and nutrition disorders) | 1 | 0
Phosphorus metabolism disorders (Metabolism and nutrition disorders) | 1 | 0
Potassium imbalance (Metabolism and nutrition disorders) | 0 | 3
Sodium imbalance (Metabolism and nutrition disorders) | 3 | 3
Total fluid volume decreased (Metabolism and nutrition disorders) | 3 | 1
Arthropathies NEC (Musculoskeletal and connective tissue disorders) | 3 | 4
Bone disorders NEC (Musculoskeletal and connective tissue disorders) | 8 | 4
Cartilage disorders (Musculoskeletal and connective tissue disorders) | 1 | 0
Fracture complications (Musculoskeletal and connective tissue disorders) | 0 | 1
Fractures NEC (Musculoskeletal and connective tissue disorders) | 1 | 0
Intervertebral disc disorders NEC (Musculoskeletal and connective tissue disorders) | 3 | 2
Joint related disorders NEC (Musculoskeletal and connective tissue disorders) | 4 | 4
Joint related signs and symptoms (Musculoskeletal and connective tissue disorders) | 4 | 6
Metabolic bone disorders (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscle infections and inflammations (Musculoskeletal and connective tissue disorders) | 2 | 0
Muscle pains (Musculoskeletal and connective tissue disorders) | 2 | 3
Muscle related signs and symptoms NEC (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscle weakness conditions (Musculoskeletal and connective tissue disorders) | 2 | 2
Musculoskeletal and connective tissue pain and discomfort (Musculoskeletal and connective tissue disorders) | 11 | 4
Myopathies (Musculoskeletal and connective tissue disorders) | 4 | 3
Osteoarthropathies (Musculoskeletal and connective tissue disorders) | 11 | 9
Rheumatoid arthropathies (Musculoskeletal and connective tissue disorders) | 0 | 1
Spine and neck deformities (Musculoskeletal and connective tissue disorders) | 7 | 5
Synovial disorders (Musculoskeletal and connective tissue disorders) | 0 | 1
Tendon disorders (Musculoskeletal and connective tissue disorders) | 0 | 5
Anal canal neoplasms malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 4
B-cell lymphomas NEC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2
Bile duct neoplasms malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Bladder neoplasms malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2
Bone neoplasms unspecified malignancy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Breast and nipple neoplasms benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Breast and nipple neoplasms malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 7 | 7
Burkitt's lymphomas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Central nervous system neoplasms malignant NEC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cervix neoplasms malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 0
Colorectal neoplasms malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 4
Endocrine neoplasms malignant and unspecified NEC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Extranodal marginal zone B-cell lymphomas (low grade B-cell) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Fallopian tube neoplasms malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Fibrous histiocytomas malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Gallbladder neoplasms malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2
Gastric neoplasms malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Glial tumours malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Gliomas benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Hepatic neoplasms malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Hodgkin's disease NEC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 2
Laryngeal neoplasms malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Leukaemias acute lymphocytic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Leukaemias chronic myeloid (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Lip and oral cavity neoplasms malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 3
Liposarcomas malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lymphomas unspecified NEC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Mediastinal neoplasms malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastases to specified sites (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 4
Myeloproliferative disorders (excl leukaemias) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Neoplasms malignant site unspecified NEC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 3
Nervous system neoplasms unspecified malignancy NEC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 5
Non-Hodgkin's lymphomas NEC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Non-small cell neoplasms malignant of the respiratory tract cell type specified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 6
Oncologic complications and emergencies (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Oropharyngeal, nasopharyngeal and tonsillar neoplasms malignant and unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Ovarian neoplasms benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Ovarian neoplasms malignant (excl germ cell) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Plasma cell myelomas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 1
Prostatic neoplasms malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 | 5
Renal neoplasms malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Renal pelvis and ureter neoplasms malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Respiratory tract and pleural neoplasms malignant cell type unspecified NEC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
Respiratory tract small cell carcinomas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Salivary gland neoplasms malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Skin melanomas (excl ocular) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Skin neoplasms benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Skin neoplasms malignant and unspecified (excl melanoma) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Soft tissue neoplasms benign NEC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Uterine neoplasms benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 5
Vulval neoplasms malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Acute polyneuropathies (Nervous system disorders) | 1 | 0
Alzheimer's disease (incl subtypes) (Nervous system disorders) | 0 | 1
Central nervous system aneurysms and dissections (Nervous system disorders) | 1 | 2
Central nervous system haemorrhages and cerebrovascular accidents (Nervous system disorders) | 5 | 9
Central nervous system vascular disorders NEC (Nervous system disorders) | 0 | 2
Cervical spinal cord and nerve root disorders (Nervous system disorders) | 1 | 0
Coordination and balance disturbances (Nervous system disorders) | 1 | 0
Cortical dysfunction NEC (Nervous system disorders) | 1 | 1
Cranial nerve disorders NEC (Nervous system disorders) | 1 | 0
Dementia (excl Alzheimer's type) (Nervous system disorders) | 1 | 0
Demyelinating disorders NEC (Nervous system disorders) | 0 | 1
Disturbances in consciousness NEC (Nervous system disorders) | 15 | 11
Encephalopathies NEC (Nervous system disorders) | 2 | 2
Encephalopathies toxic and metabolic (Nervous system disorders) | 0 | 1
Facial cranial nerve disorders (Nervous system disorders) | 1 | 0
Generalised tonic-clonic seizures (Nervous system disorders) | 1 | 0
Headaches NEC (Nervous system disorders) | 6 | 3
Hydrocephalic conditions (Nervous system disorders) | 1 | 1
Increased intracranial pressure disorders (Nervous system disorders) | 1 | 1
Lumbar spinal cord and nerve root disorders (Nervous system disorders) | 2 | 1
Memory loss (excl dementia) (Nervous system disorders) | 2 | 0
Migraine headaches (Nervous system disorders) | 1 | 1
Mononeuropathies (Nervous system disorders) | 3 | 1
Motor neurone diseases (Nervous system disorders) | 0 | 1
Nervous system disorders NEC (Nervous system disorders) | 1 | 0
Neurological signs and symptoms NEC (Nervous system disorders) | 10 | 4
Neuromuscular disorders NEC (Nervous system disorders) | 0 | 1
Optic nerve disorders NEC (Nervous system disorders) | 0 | 1
Paraesthesias and dysaesthesias (Nervous system disorders) | 3 | 1
Paralysis and paresis (excl cranial nerve) (Nervous system disorders) | 5 | 1
Parkinson's disease and parkinsonism (Nervous system disorders) | 1 | 1
Peripheral neuropathies NEC (Nervous system disorders) | 2 | 1
Seizures and seizure disorders NEC (Nervous system disorders) | 9 | 14
Speech and language abnormalities (Nervous system disorders) | 1 | 0
Spinal cord and nerve root disorders NEC (Nervous system disorders) | 4 | 4
Structural brain disorders NEC (Nervous system disorders) | 1 | 2
Transient cerebrovascular events (Nervous system disorders) | 3 | 4
Abortions spontaneous (Pregnancy, puerperium and perinatal conditions) | 1 | 0
Device issues NEC (Product Issues) | 1 | 0
Abnormal behaviour NEC (Psychiatric disorders) | 1 | 0
Anxiety symptoms (Psychiatric disorders) | 2 | 0
Behaviour and socialisation disturbances (Psychiatric disorders) | 1 | 0
Bipolar disorders (Psychiatric disorders) | 2 | 2
Confusion and disorientation (Psychiatric disorders) | 1 | 2
Deliria (Psychiatric disorders) | 0 | 1
Delusional disorders (Psychiatric disorders) | 0 | 1
Delusional symptoms (Psychiatric disorders) | 1 | 0
Depressive disorders (Psychiatric disorders) | 6 | 10
Mental disorders NEC (Psychiatric disorders) | 10 | 6
Mood alterations with manic symptoms (Psychiatric disorders) | 1 | 1
Mood disorders NEC (Psychiatric disorders) | 0 | 2
Panic attacks and disorders (Psychiatric disorders) | 1 | 0
Psychotic disorder NEC (Psychiatric disorders) | 8 | 6
Schizoaffective and schizophreniform disorders (Psychiatric disorders) | 1 | 2
Schizophrenia NEC (Psychiatric disorders) | 1 | 4
Somatic symptom disorders (Psychiatric disorders) | 3 | 0
Substance related and addictive disorders (Psychiatric disorders) | 9 | 4
Suicidal and self-injurious behaviour (Psychiatric disorders) | 33 | 28
Bladder disorders NEC (Renal and urinary disorders) | 0 | 1
Genital and urinary tract disorders NEC (Renal and urinary disorders) | 2 | 3
Glomerulonephritis and nephrotic syndrome (Renal and urinary disorders) | 0 | 1
Nephropathies and tubular disorders NEC (Renal and urinary disorders) | 1 | 0
Renal failure and impairment (Renal and urinary disorders) | 25 | 24
Renal lithiasis (Renal and urinary disorders) | 4 | 4
Renal obstructive disorders (Renal and urinary disorders) | 0 | 1
Renal vascular and ischaemic conditions (Renal and urinary disorders) | 0 | 1
Structural and obstructive urethral disorders (excl congenital) (Renal and urinary disorders) | 1 | 0
Urethral disorders NEC (Renal and urinary disorders) | 0 | 1
Urinary abnormalities (Renal and urinary disorders) | 0 | 2
Urinary tract lithiasis NEC (Renal and urinary disorders) | 3 | 2
Urinary tract signs and symptoms NEC (Renal and urinary disorders) | 1 | 0
Breast disorders NEC (Reproductive system and breast disorders) | 1 | 1
Cervix disorders NEC (Reproductive system and breast disorders) | 3 | 3
Menstruation and uterine bleeding NEC (Reproductive system and breast disorders) | 1 | 0
Menstruation with increased bleeding (Reproductive system and breast disorders) | 4 | 2
Ovarian and fallopian tube cysts and neoplasms (Reproductive system and breast disorders) | 2 | 1
Pelvis and broad ligament disorders NEC (Reproductive system and breast disorders) | 1 | 0
Prostate and seminal vesicles infections and inflammations (Reproductive system and breast disorders) | 0 | 2
Prostatic neoplasms and hypertrophy (Reproductive system and breast disorders) | 2 | 1
Reproductive tract disorders NEC (excl neoplasms) (Reproductive system and breast disorders) | 0 | 1
Testicular and epididymal disorders NEC (Reproductive system and breast disorders) | 1 | 0
Uterine disorders NEC (Reproductive system and breast disorders) | 2 | 0
Vulvovaginal disorders NEC (Reproductive system and breast disorders) | 0 | 2
Breathing abnormalities (Respiratory, thoracic and mediastinal disorders) | 12 | 9
Bronchial conditions NEC (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Bronchospasm and obstruction (Respiratory, thoracic and mediastinal disorders) | 30 | 22
Conditions associated with abnormal gas exchange (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Coughing and associated symptoms (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Laryngeal and adjacent sites disorders NEC (excl infections and neoplasms) (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Lower respiratory tract signs and symptoms (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Mediastinal disorders (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Nasal disorders NEC (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Parenchymal lung disorders NEC (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Pneumothorax and pleural effusions NEC (Respiratory, thoracic and mediastinal disorders) | 7 | 4
Pulmonary hypertensions (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary oedemas (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Pulmonary thrombotic and embolic conditions (Respiratory, thoracic and mediastinal disorders) | 11 | 21
Respiratory failures (excl neonatal) (Respiratory, thoracic and mediastinal disorders) | 6 | 6
Respiratory tract disorders NEC (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Angioedemas (Skin and subcutaneous tissue disorders) | 3 | 2
Dermatitis and eczema (Skin and subcutaneous tissue disorders) | 2 | 2
Dermatitis ascribed to specific agent (Skin and subcutaneous tissue disorders) | 0 | 1
Lipodystrophies (Skin and subcutaneous tissue disorders) | 1 | 0
Pruritus NEC (Skin and subcutaneous tissue disorders) | 1 | 0
Psoriatic conditions (Skin and subcutaneous tissue disorders) | 0 | 1
Rashes, eruptions and exanthems NEC (Skin and subcutaneous tissue disorders) | 0 | 1
Skin and subcutaneous tissue ulcerations (Skin and subcutaneous tissue disorders) | 1 | 3
Criminal activity (Social circumstances) | 1 | 0
Abdominal therapeutic procedures NEC (Surgical and medical procedures) | 0 | 1
Biliary tract and gallbladder therapeutic procedures (Surgical and medical procedures) | 0 | 1
Cardiac therapeutic procedures NEC (Surgical and medical procedures) | 1 | 0
Cardiac valve therapeutic procedures (Surgical and medical procedures) | 0 | 2
Facial therapeutic procedures (Surgical and medical procedures) | 0 | 1
Gastric therapeutic procedures (Surgical and medical procedures) | 1 | 1
Hernia repairs (Surgical and medical procedures) | 1 | 2
Joint therapeutic procedures (Surgical and medical procedures) | 2 | 3
Laryngeal therapeutic procedures (Surgical and medical procedures) | 0 | 1
Limb therapeutic procedures (Surgical and medical procedures) | 2 | 0
Penile therapeutic procedures (Surgical and medical procedures) | 0 | 1
Psychiatric therapies (Surgical and medical procedures) | 1 | 0
Renal therapeutic procedures (Surgical and medical procedures) | 1 | 0
Small intestine therapeutic procedures (Surgical and medical procedures) | 1 | 0
Soft tissue therapeutic procedures NEC (Surgical and medical procedures) | 0 | 1
Spine and spinal cord therapeutic procedures (Surgical and medical procedures) | 2 | 3
Therapeutic procedures NEC (Surgical and medical procedures) | 1 | 2
Uterine therapeutic procedures (Surgical and medical procedures) | 1 | 1
Accelerated and malignant hypertension (Vascular disorders) | 0 | 1
Aortic aneurysms and dissections (Vascular disorders) | 0 | 1
Aortic embolism and thrombosis (Vascular disorders) | 0 | 1
Circulatory collapse and shock (Vascular disorders) | 0 | 2
Haemorrhages NEC (Vascular disorders) | 2 | 2
Lymphoedemas (Vascular disorders) | 1 | 0
Non-site specific embolism and thrombosis (Vascular disorders) | 2 | 1
Non-site specific necrosis and vascular insufficiency NEC (Vascular disorders) | 1 | 0
Peripheral embolism and thrombosis (Vascular disorders) | 9 | 11
Peripheral vasoconstriction, necrosis and vascular insufficiency (Vascular disorders) | 1 | 1
Varicose veins NEC (Vascular disorders) | 0 | 1
Vascular hypertensive disorders NEC (Vascular disorders) | 6 | 7
Vascular hypotensive disorders (Vascular disorders) | 3 | 4
Vasculitides NEC (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Pitavastatin (N=3888) | Placebo (N=3881)
Physical examination procedures and organ system status (Investigations) | 62 | 65
Renal function analyses (Investigations) | 125 | 122
Diabetes mellitus (incl subtypes) (Metabolism and nutrition disorders) | 238 | 184
General nutritional disorders NEC (Metabolism and nutrition disorders) | 66 | 44
Muscle pains (Musculoskeletal and connective tissue disorders) | 77 | 44
Musculoskeletal and connective tissue pain and discomfort (Musculoskeletal and connective tissue disorders) | 40 | 43
Vascular hypertensive disorders NEC (Vascular disorders) | 37 | 50

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (4):
  • Study Protocol and Informed Consent Form: English (2022-05-16): https://cdn.clinicaltrials.gov/large-docs/90/NCT02344290/Prot_ICF_003.pdf
  • Statistical Analysis Plan: REPRIEVE SAP (2022-06-06): https://cdn.clinicaltrials.gov/large-docs/90/NCT02344290/SAP_004.pdf
  • Statistical Analysis Plan: Mechanistic Substudy SAP (2023-10-04): https://cdn.clinicaltrials.gov/large-docs/90/NCT02344290/SAP_005.pdf
  • Informed Consent Form: Spanish (2022-05-16): https://cdn.clinicaltrials.gov/large-docs/90/NCT02344290/ICF_006.pdf